# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

**DMID Protocol: 20-0006** 

**Study Title:** 

A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Adults (ACTT-2)

NC04280705

**ACTT-2 Version 3.0** 

**DATE: 20-AUG-2020** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

# **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 20-0006 (ACTT-2) |
|---|---|
| <b>Development Phase:</b> | Phase 3 |
| Products: | Baricitinib + Remdesivir |
| | Remdesivir |
| Form/Route: | IV (Remdesivir) and PO (Baricitinib/Placebo) |
| Indication Studied: | COVID-19 |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | May 8, 2020 |
| Clinical Trial Completion Date: | Trial Ongoing |
| Date of the Analysis Plan: | August 20, 2020 |
| Version Number: | 3.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | II |
|---|---|---|
| TABLE | OF CONTENTS | III |
| LIST OF | ABBREVIATIONS | VI |
| 1. | PREFACE | 8 |
| 2. | INTRODUCTION | 9 |
| 2.1. | Purpose of the Analyses | 9 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 11 |
| 3.1. | Study Objectives | 11 |
| 3.2. | Endpoints | 12 |
| 3.3. | Study Definitions and Derived Variables | 13 |
| 3.3.1. | Baseline Value | 13 |
| 3.3.2. | Recovery and Time to Recovery | 13 |
| 3.3.3. | Clinical Status at Specific Timepoints | 14 |
| 3.3.4. | Time to Clinical Status Improvement | 14 |
| 3.3.5. | Time to Discharge or NEWS of ≤ 2 | 15 |
| 3.3.6. | Days of Non-invasive ventilation/high-flow oxygen | 15 |
| 3.3.7. | Days of Invasive Mechanical Ventilation/ECMO | |
| 3.3.8. | Days of Oxygen | 15 |
| 3.3.9. | Days of Hospitalization | 16 |
| 3.3.10. | Time to Death | 16 |
| 3.3.11. | Composite Endpoint of Death, SAEs, Severe AEs, Discontinuation of Study Product Administrations | 16 |
| 4. | INVESTIGATIONAL PLAN | 17 |
| 4.1. | Overall Study Design and Plan | 17 |
| 4.2. | Selection of Study Population | 17 |
| 4.2.1. | Treatments Administered. | |
| 4.2.2. | Identity of Investigational Product(s) | 17 |
| 4.2.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 17 |
| 4.2.4. | Selection of Doses in the Study | 18 |
| 4.2.5. | Selection and Timing of Dose for Each Subject | |
| 4.2.6. | Blinding | 18 |

# **Table of Contents** (continued)

| 4.2.7. | Prior and Concomitant Therapy | 18 |
|--------|--------------------------------------------------------|----|
| 4.2.8. | Treatment Compliance | 18 |
| 4.3. | Efficacy and Safety Variables | 18 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 21 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 22 |
| 6.1. | General Principles | 22 |
| 6.2. | Timing of Analyses | 23 |
| 6.2.1. | Early Sample Size Reassessment | 23 |
| 6.2.2. | Interim analyses | 23 |
| 6.2.3. | Final Analyses | 23 |
| 6.3. | Analysis Populations | 23 |
| 6.3.1. | Intention-to-Treat (ITT) and As Treated Populations | 23 |
| 6.4. | Covariates and Subgroups | 24 |
| 6.5. | Missing Data | 26 |
| 6.6. | Interim Analyses and Data Monitoring | 27 |
| 6.6.1. | Interim Safety Analyses | 27 |
| 6.6.2. | Interim Efficacy Review | 27 |
| 6.7. | Multicenter Studies | 28 |
| 6.8. | Multiple Comparisons/Multiplicity | 28 |
| 7. | STUDY SUBJECTS | 29 |
| 7.1. | Disposition of Subjects | 29 |
| 7.2. | Protocol Deviations | 29 |
| 8. | EFFICACY EVALUATION | 30 |
| 8.1. | Primary Efficacy Analysis | 30 |
| 8.1.1. | Primary Analyses | 30 |
| 8.1.2. | Supplemental and Sensitivity Analyses | 31 |
| 8.2. | Secondary Efficacy Analyses | 32 |
| 8.2.1. | Ordinal Scale Outcomes (Key Secondary Outcome Measure) | 32 |
| 8.2.2. | NEWS | 33 |
| 8.2.3. | Days of Oxygenation | 33 |
| 8.2.4. | Incidence of New Oxygen use | 34 |

# **Table of Contents** (continued)

| 8.2.5. | Days of Non-Invasive Ventilation/High-Flow Oxygen | 34 |
|---|---|---|
| 8.2.6. | Incidence of New Non-Invasive Ventilation/High-Flow Oxygen | |
| 8.2.7. | Days of Invasive Mechanical Ventilation/ECMO | |
| 8.2.8. | Incidence of New Invasive Mechanical Ventilation/ECMO | |
| 8.2.9. | Days of Hospitalization | |
| 8.3. | Exploratory Efficacy Analyses | |
| 9. | SAFETY EVALUATION | |
| 9.1. | Demographic and Other Baseline Characteristics | 35 |
| 9.1.1. | Prior and Concurrent Medical Conditions | |
| 9.1.2. | Prior and Concomitant Medications | 35 |
| 9.2. | Measurements of Treatment Compliance | 36 |
| 9.3. | Adverse Events | |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 36 |
| 9.5. | Pregnancies | 37 |
| 9.6. | Clinical Laboratory Evaluations | 38 |
| 9.7. | Vital Signs and Physical Evaluations | 38 |
| 9.8. | Concomitant Medications | 38 |
| 9.9. | Other Safety Measures | 38 |
| 10. | PHARMACOKINETICS | 39 |
| 11. | IMMUNOGENICITY | 40 |
| 12. | OTHER ANALYSES | 41 |
| 13. | REPORTING CONVENTIONS | 42 |
| 14. | TECHNICAL DETAILS | 43 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 44 |
| 16. | REFERENCES | 48 |
| 17. | LISTING OF TABLES, FIGURES, AND LISTINGS | 49 |
| APPENI | DIX 1. TABLE MOCK-UPS | |
| APPENI | DIX 2. FIGURE MOCK-UPS | 101 |
| A DDENII | OIY 3 LISTINGS MOCK-HPS | 124 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|------------|--------------------------------------------------|
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| BEEC | Blinded Endpoint Evaluation Committee |
| CI | Confidence Interval |
| CoV / COV | Coronavirus |
| CRF / eCRF | Case Report Form / Electronic Case Report Form |
| CSR | Clinical Study Report |
| DAIDS | Division of AIDS |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| ECMO | Extracorporeal Membrane Oxygenation |
| FDA | Food and Drug Administration |
| GMT | Geometric Mean Titer |
| GMFR | Geometric Mean Fold Rise |
| ICH | International Conference on Harmonisation |
| ITT | Intention to Treat |
| IV | Intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| MOP | Manual of Procedures |
| N | Number (typically refers to subjects) |
| NEWS | National Early Warning Score |
| NIH | National Institutes of Health |
| OP | Oropharyngeal |
| PCR | Polymerase Chain Reaction |
| PI | Principal Investigator |
| PT | Preferred Term / Prothrombin Time |
| RCD | Reverse Cumulative Distribution |
| RDV | Remdesivir |

| RNA | Ribonucleic Acid |
|------|------------------------------------------|
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SARS | Severe Acute Respiratory Syndrome |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SOC | System Organ Class |
| US | United States |
| WBC | White Blood Cell |
| WHO | World Health Organization |

# 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Adults" (DMID Protocol 20-0006) describes and expands upon the statistical information presented in the protocol. This protocol is an adaptive protocol with different stages. Each stage will have a separate SAP. This SAP is for the study's 2<sup>nd</sup> stage "ACTT-2": Baricitinib + Remdesivir vs. Remdesivir.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA) and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains: a review of the study design, general statistical considerations, comprehensive statistical analysis methods for efficacy and safety outcomes, and a list of proposed tables, figures and listings. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

# 2. INTRODUCTION

A preliminary review of data from ACTT-1 occurring after 606 recoveries and 103 deaths (approximately 67% of the 1063 subjects enrolled) demonstrated that subjects that received remdesivir had a 31% faster time to recovery (11 vs 15 days, recovery rate ratio 1.312 (1.119, 1.541), p<0.001), and a decrease in mortality (8.0% vs 11.6%, p = 0.059). The Data and Safety Monitoring Board (DSMB) asked that the sponsor be unblinded early given public health implications and implications for ACTT-2. While an antiviral appears to have some efficacy in the treatment of COVID-19, the mortality rate is still high. Infection by pathogenic coronaviruses (e.g. SARS and SARS-CoV-2) often results in excessive cytokine and chemokine action with the development of acute respiratory distress syndrome (ARDS). It is postulated that this dysregulated inflammatory immune response is contributing to the excessive mortality and targeting this response will further improve outcomes.

Baricitinib, an orally administered, selective inhibitor of Janus Kinase (JAK)1 and JAK2, could be a therapeutic option because of the potential to inhibit signaling from multiple cytokines in COVID-19 patients. Baricitinib inhibits signaling of cytokines implicated in COVID-19, including interleukin (IL) IL-2, IL-6, IL-10, Interferon gamma (IFN-γ), and Granulocyte colony-stimulating factor (G-CSF), with lower IC<sub>50</sub> values translating to a greater overall inhibition of STAT signaling during the dosing interval. Baricitinib treatment resulted in a reduction from baseline in serum IL-6 at Week 12 in patients with active rheumatoid arthritis (RA) in a Phase 2, randomized, placebo-controlled study of baricitinib (data on file). The potent anti-inflammatory effects of baricitinib have also been demonstrated by the reduction of serum levels of IFN-γ, IP-10, Granulocyte-macrophage colony-stimulating factor (GM-CSF) and monocyte chemoattractant protein (MCP-1) in pediatric patients with steroid-dependent chronic inflammation, resulting in control of disease activity and the ability to wean or taper steroids.

Baricitinib is already approved for treatment of rheumatoid arthritis. It is administered orally once a day, with good oral bioavailability. It has a short half-life (approximately 12 hours in RA patients), so treatment can be interrupted or stopped if necessary. It has few drug-drug interactions (due to low CYP inhibitory activity) so it can be given concomitantly with background therapies. Baricitinib has a well-established safety profile, based on clinical trial data and post-marketing data in patients with RA. This profile, together with the observation that baricitinib is a potent AAK1/BIKE/GAK inhibitor with known anti-cytokine effects, provide the rationale to study baricitinib in the context of a randomized, controlled clinical trial in patients with COVID-19.

# 2.1. Purpose of the Analyses

This SAP encompasses all interim analyses and the final analysis of primary and secondary outcome measures. These analyses will assess the efficacy and safety of baricitinib + remdesivir in comparison with remdesivir and will be included in the Clinical Study Report. This protocol is an adaptive design and, if the design is modified, the SAP will be amended accordingly. The protocol for DMID 20-0006 calls for a planned interim efficacy analysis once roughly 33% of the targeted number of recoveries have been observed, and ongoing safety analyses. Safety interim analyses occur more frequently to review safety data in the event that the experimental agent inflicts harm. The goal of the efficacy interim analyses is to review endpoint data in order

to recommend whether the current study arm should proceed or to stop early for benefit or futility.

This SAP describes the planned analysis to be conducted by the Investigational New Drug (IND) sponsor NIAID. Additionally, there will be a separate analysis by the Manufacturer, Lilly USA, in which Lilly will:

- Define key secondary endpoints that will be tested with adjustments for multiple comparison. The adjustment is through a graphical testing scheme that controls for family-wise type I error;
- Pre-specify details of handling of intercurrent events including imputation procedures;
- Define additional analysis of time-to-event data that account for competing risk;
- Define additional safety analysis will also be pre-specified in the Addendum SAP

These analyses are useful to the manufacturer for regulatory purposes and will be pre-specified in an Addendum to this SAP.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

# **Primary Objective**

To evaluate the clinical efficacy, as assessed by time to recovery, of different investigational therapeutics as compared to the control arm.

# **Secondary Objectives**

The key secondary objective is to evaluate the clinical efficacy of different investigational therapeutics relative to the control arm in adults hospitalized with COVID-19 according to clinical status (8-point ordinal clinical scale) at Day 15.

The other secondary objectives are to:

- 1. Evaluate clinical efficacy of different investigational therapeutics as compared to the control arm as assessed by:
  - Clinical Severity
    - o 8-Point Clinical Status Ordinal scale:
      - Time to an improvement of one category and two categories from Day 1 (baseline) on the clinical status 8-point ordinal scale.
      - Subject clinical status using 8-point ordinal scale at Days 3, 5, 8, 11, 15, 22, and 29.
      - Mean change in the clinical status 8-point ordinal scale from Day 1 to Days 3, 5, 8, 11, 15, and 29.
    - o National Early Warning Score (NEWS):
      - Time to discharge or to a NEWS of  $\leq$  2 and maintained for 24 hours, whichever occurs first.
      - Change from Day 1 to Days 3, 5, 8, 11, 15, and 29 in NEWS.
    - o Oxygenation:
      - Oxygenation use up to Day 29.
      - Incidence and duration of new oxygen use through Day 29.
    - o Non-invasive ventilation/high flow oxygen:
      - Non-invasive ventilation/high flow oxygen use up to Day 29.
      - Incidence and duration of new non-invasive ventilation or high flow oxygen use through Day 29.
    - o Invasive Mechanical Ventilation / extracorporeal membrane oxygenation (ECMO):
      - Ventilator/ECMO use up to Day 29.
      - Incidence and duration of new mechanical ventilation or ECMO use through Day 29.

- Hospitalization
  - o Duration of hospitalization (in days) through Day 29.
- Mortality
  - o 14-day mortality.
  - o 28-day mortality.
- 2. Evaluate the safety of the intervention through 28 days of follow-up as compared to the control arm as assessed by:
  - Cumulative incidence of SAEs through Day 29
  - Cumulative incidence of Grade 3 and 4 clinical and/or laboratory AEs through Day 29.
  - Discontinuation or temporary suspension of study product administrations (for any reason).
  - Changes in white cell count (WBC) with differential, hemoglobin, platelets, creatinine, glucose, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and prothrombin time (PT reported as INR), d-dimer, and C-reactive protein (CRP) over time (analysis of lab values in addition to AEs noted above).

# **Exploratory Objective**

The exploratory objective is to evaluate the virologic efficacy of different investigational therapeutics as compared to the control arm as assessed by:

- Percentage of subjects with SARS-CoV-2 detectable in oropharyngeal (OP) sample at Day 3, 5, 8, 11, 15, and 29.
- Quantitative SARS-CoV-2 virus in OP sample at Day 3, 5, 8, 11, 15, and 29.
- Development of resistance of SARS-CoV-2 in OP sample at Day 3, 5, 8, 11, 15, and 29.
- Quantitative SARS-CoV-2 virus in blood at Day 3, 5, 8, and 11.

# 3.2. Endpoints

#### **Primary Endpoint**

Time to recovery, where recovery is defined as clinical status in states 1, 2, or 3 of the 8-point ordinal scale, censored at Day 29.

- Clinical status of a subject (8-point ordinal scale) is defined below:
  - 8. Death;
  - 7. Hospitalized, on invasive mechanical ventilation or ECMO;
  - 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  - 5. Hospitalized, requiring supplemental oxygen;
  - 4. Hospitalized, not requiring supplemental oxygen requiring ongoing medical care (COVID-19 related or otherwise);

- 3. Hospitalized, not requiring supplemental oxygen no longer requiring ongoing medical care;
- 2. Not hospitalized, limitation on activities and/or requiring home oxygen;
- 1. Not hospitalized, no limitations on activities

# **Secondary Endpoints**

The key secondary endpoint is clinical status (8-point ordinal scale) on Day 15.

The other secondary endpoints are:

- Ordinal outcome assessed daily while hospitalized and on Days 15, 22, and 29.
- NEWS assessed daily while hospitalized and on Days 15 and 29.
- Days of supplemental oxygen (if applicable).
- Days of non-invasive ventilation/high-flow oxygen (if applicable).
- Days of invasive mechanical ventilation/ECMO (if applicable).
- Days of hospitalization.
- Date and cause of death (if applicable).
- SAEs.
- Grade 3 and 4 adverse events
- WBC with differentials, hemoglobin, platelets, creatinine, glucose, total bilirubin, ALT, AST, INR, d-dimer, and CRP on Day 1; Days 3, 5, 8, and 11 (while hospitalized); and Days 15 and 29 (if attends in-person visit or still hospitalized).

#### **Exploratory Endpoint**

- Qualitative and quantitative polymerase chain reaction PCR for SARS-CoV-2 in OP swab on Day 1; Days 3, 5, 8, and 11 (while hospitalized); and Days 15 and 29 (if attends in-person visit or still hospitalized).
- Qualitative and quantitative PCR for SARS-CoV-2 in blood on Day 1; Days 3, 5, 8, and 11 (while hospitalized).

# 3.3. Study Definitions and Derived Variables

#### 3.3.1. Baseline Value

For efficacy assessments, the baseline value will be defined as the last value obtained prior to randomization. For safety assessments, the baseline value will be defined as the last value obtained prior to the first dose of study product on trial.

#### 3.3.2. Recovery and Time to Recovery

The primary efficacy outcome measure is the time to recovery. Recovery will be defined as having a value of 1, 2, or 3 on the clinical status 8-point ordinal scale. The time to recovery will be defined as the elapsed time (in days) from randomization to the earliest day at which a subject

reaches recovery. Note that since clinical status assessments are recorded as defined in Section 4.3, the day that is being assessed (not necessarily the day the response is collected) will be used to determine the timing of events. For example, a subject with a score of 5 recorded on Days 1 - 3 and a score of 3 recorded on Day 4 will have a time to recovery equal to 3 days. It is also possible that a subject has a clinical status score > 3 reported for a particular day but was subsequently discharged on the same day. Such cases will be reviewed by the NIAID Medical Officer to make the determination of whether the subject should be considered recovered in analyses. Subject data to be reviewed as part of this determination will include the reported clinical status scores while hospitalized, where the subject was discharged to (e.g. private residence, rehabilitation facility, long-term care/nursing home), and any information regarding readmittance.

Any subjects that are lost to follow-up or terminated early prior to an observed recovery will be censored at the day of their last observed assessment. Subjects who complete follow-up but do not experience recovery will be censored at the day of their Day 29 visit. All deaths within Day 29 (and prior to recovery) will be considered censored at 28 days. Note that we do not expect many subjects to worsen after discharge.

However, we will evaluate whether any discharged subjects subsequently experience a worse clinical status and sensitivity analyses will be conducted accordingly. For these analyses, subjects who recover but are later re-admitted for COVID-19 will not be considered a recovery but will instead be censored at 28 days.

# 3.3.3. Clinical Status at Specific Timepoints

The key secondary analyses include evaluation of the clinical status score at Day 15. For this outcome, Study Visit Day 15 is the timepoint of interest, not necessarily the actual study day. The score collected at the study visit corresponding to Day 15 will be used for this outcome. For analyses of this outcome, imputation of the clinical score may be performed following the rules described in Section 6.5.

Additional analyses are clinical status at Days 3, 5, 8, 11, 15, 22, and 29. As the with above, the scores that will be used are those collected at the study visits corresponding to those days.

#### 3.3.4. Time to Clinical Status Improvement

Additional analyses will evaluate the time to improvement of at least one point on the clinical status 8-point ordinal scale. That is, improvement will be defined as a decrease of at least one point on the 8-point scale compared to the baseline value (e.g. from 5 to 4; from 5 to 3) and the time to improvement will be defined as the elapsed time (in days) from randomization to the earliest day of observed improvement. Note that since clinical status assessments are recorded as defined in Section 4.3, the day that is being assessed (not necessarily the day the response is collected) will be used to determine the timing of events.

For analyses of this outcome, imputation of the clinical score may be performed following the rules described in Section 6.5.

Any subjects that are lost to follow-up or terminated early prior to an observed improvement will be censored at the day of their last observed assessment. Subjects who complete follow-up but do

not experience improvement will be censored at the day of their Day 29 visit. All deaths within Day 29 (and prior to improvement) will be considered censored at 28 days.

An alternative definition of improvement will also be used where improvement will be defined as a decrease of at least two points on the 8-point scale compared to the baseline value (e.g. from 5 to 3; from 5 to 2). The timing and censoring definitions will follow similarly to the above.

# 3.3.5. Time to Discharge or NEWS of $\leq 2$

The time to discharge or NEWS of  $\leq 2$  will be defined as the elapsed time (in days) from baseline to the earliest day at which either of the following occur:

- Discharge from hospital
- Reported NEWS of  $\leq 2$  which is maintained for 24 hours

For the latter bullet, to meet this criterion, scores of  $\leq 2$  must be reported on consecutive study visits. The timing of the event will be set to the day of the second assessment.

All deaths that occur before discharge or before an observed NEWS of  $\leq$  2 will be considered censored at 28 days.

# 3.3.6. Days of Non-invasive ventilation/high-flow oxygen

Non-invasive ventilation/high flow-oxygen days will be defined as the number of days where the clinical status score is equal to 6. After discharge, the Post-Discharge Supplemental Oxygen CRF questions regarding days of non-invasive ventilation or high-flow oxygen will be used. The total number of days will be the sum of all reported days, regardless of whether the days occur consecutively or in disjoint intervals. See Section 6.5 for the plan for handling subjects who do not have data through Day 29 or die prior to Day 29.

#### 3.3.7. Days of Invasive Mechanical Ventilation/ECMO

Invasive Mechanical Ventilator / ECMO days will be defined as the number of days where the clinical status score is equal to 7. After discharge, the Post-Discharge Supplemental Oxygen CRF questions regarding days of ECMO or invasive ventilation will be used. The total number of days will be the sum of all reported days, regardless of whether the days occur consecutively or in disjoint intervals. See Section 6.5 for the plan for handling subjects who do not have data through Day 29 or die prior to Day 29.

# 3.3.8. Days of Oxygen

Oxygen days will be defined as the number of days where the clinical status score is equal to 5, 6, or 7. After discharge, the Post-Discharge Supplemental Oxygen CRF question regarding days of oxygenation (including ECMO, invasive ventilation, non-invasive ventilation, high-flow oxygen devices, and all other oxygen delivery devices) will be used. The total number of days will be the sum of all reported days, regardless of whether the days occur consecutively or in disjoint intervals. See Section 6.5 for the plan for handling subjects who do not have data through Day 29 or die prior to Day 29.

# 3.3.9. Days of Hospitalization

Duration (in days) of hospitalization will be defined as the number of days subject is hospitalized for COVID-19-related reasons starting from the date of randomization. It will be calculated as the total number of days hospitalized, including readmissions for COVID-19-related reason. See Section 6.5 for the plan for handling subjects who do not have data through Day 29 or die prior to Day 29.

#### 3.3.10. Time to Death

For analysis of time to death, the time to death will be defined as the elapsed time (in days) from randomization (or treatment administration for the safety analysis) to death. Any subjects that are lost to follow-up or terminated early prior to death will be censored at the day of their last observed assessment or last captured event (e.g. the end date of an adverse event). If it is learned that a subject who terminated early had subsequently died prior to Day 29, then the subject will be classified as dead. Subjects who complete follow-up will be censored at the earliest of their Day 29 visit and (actual) Day 29. Deaths that occur after Day 29 will be censored at Day 29.

Similar censoring methods will be used for the 14-day mortality analyses in that deaths that occur after Day 15 will be censored at Day 15 and subjects who are confirmed alive through Day 15 will be censored at Day 15. Subjects whose last observed assessment or last capture event (e.g. the end date of an adverse event) is prior to Day 15 will be censored at that last observed assessment/event.

# 3.3.11. Composite Endpoint of Death, SAEs, Severe AEs, Discontinuation of Study Product Administrations

A safety composite endpoint will be defined as the occurrence of at least one of the following through Day 29:

- 1. Death
- 2. SAE
- 3. Grade 3 or 4 AE

The time to this composite endpoint will be defined as the elapsed time (in days) from baseline to the earliest date of any of the events. Any subjects that are lost to follow-up or terminated early prior to experiencing any of the events will be censored at the day of their last observed assessment. Subjects who complete follow-up but do not experience any of the events will be censored at the Day 29 visit.

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

ACTT-2 will evaluate the combination of baricitinib and remdesivir compared to remdesivir alone. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests and OP swab and blood (serum only) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the subject to return to the clinic. In this case, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone.

# 4.2. Selection of Study Population

Male and non-pregnant female adults  $\geq$ 18 years of age or older with COVID-19 and who meet all eligibility criteria will be enrolled at up to approximately 100 clinical trial sites globally. The target population should reflect the community at large.

See Section 5.1 and 5.2 of Appendix B of the study protocol for the full list of inclusion and exclusion criteria.

#### 4.2.1. Treatments Administered

All subjects will receive remdesivir as a 200 mg intravenous (IV) loading dose on Day 1, followed by a 100 mg once-daily IV maintenance dose for the duration of the hospitalization up to a 10-day total course.

For the baricitinib component, subjects will receive either active product or placebo as follows:

- Baricitinib will be administered as a 4 mg orally (po) (two 2mg tablets) or crushed for NG tube, daily for the duration of the hospitalization up to a 14-day total course.
- A placebo will be given as two tablets po or crushed for NG tube, daily for the duration of the hospitalization up to a 14-day total course.

# 4.2.2. Identity of Investigational Product(s)

See Section 6.1.1 of Appendix B of the study protocol.

# 4.2.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment and randomization of subjects is done online using the enrollment module of Advantage eClinical<sup>®</sup>.

Eligible subjects will be randomized and assigned in a 1:1 ratio to either baricitinib + remdesivir or remdesivir, with stratification by site and disease severity by ordinal scale (Moderate disease [4 or 5 on the ordinal scale]) or Severe disease [6 or 7 on the ordinal scale]). The randomization is based on a variable blocked scheme to provide an approximately balanced allocation to the treatment groups during the study. If arms are added or removed later in the study, randomization will continue in an equal allocation manner.

## 4.2.4. Selection of Doses in the Study

The dose of remdesivir used in this study will be the same dose that has been used in the human Ebola clinical trials.

# 4.2.5. Selection and Timing of Dose for Each Subject

See Sections 6.1.2 through 6.1.5 of Appendix B of the study protocol.

# 4.2.6. Blinding

As both arms are receiving remdesivir, the remdesivir product is not blinded and study infusions can be labeled accordingly.

The baricitinib/placebo component is blinded. Baricitinib and placebo tablets are identical in appearance.

Unblinding of the study will occur after all subjects enrolled have reached the end of study, and these visits are monitored and data is cleaned, or if the DSMB recommends unblinding.

If AEs occur and investigators are concerned about the treatment allocation, the treatment can be discontinued. If a Serious Adverse Event occurs, that is thought to be related to the study drug, and the treating clinician believes that knowledge of the treatment arm may change the therapy provided to the patient, the individual subject can be unblinded. The procedure for unblinding will be further detailed in the Manual of Procedures (MOP).

# 4.2.7. Prior and Concomitant Therapy

See Section 6.5.1 of Appendix B of the study protocol for permitted concomitant therapy and procedures. See Section 6.5.2 of Appendix B of the study protocol for prohibited concomitant therapies.

#### 4.2.8. Treatment Compliance

See Section 6.1.4 of Appendix B of the study protocol for details on dose modifications.

Each dose of study product will be administered by a member of the clinical research team who is qualified and licensed to administer the study product. Administration and date, and time, will be entered into the case report form (CRF).

# 4.3. Efficacy and Safety Variables

For each study day while the patient is hospitalized, the clinical status will be recorded on an 8-point ordinal scale as follows:

- Day 1 The clinical assessment at the time of randomization.
- Day 2 + The most severe assessment occurring from midnight to midnight (00:00 to 23:59) of the prior day (e.g., the value recorded on Day 3 will be the most severe outcome that occurred on Day 2).

where the clinical status scale is defined as follows:

8. Death;

- 7. Hospitalized, on invasive mechanical ventilation or ECMO;
- 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
- 5. Hospitalized, requiring supplemental oxygen;
- 4. Hospitalized, not requiring supplemental oxygen- requiring ongoing medical care (COVID-19 related or otherwise);
- 3. Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care:
- 2. Not hospitalized, limitation on activities;
- 1. Not hospitalized, no limitations on activities

A modified version of the ordinal scale will be used in sensitivity analyses of the primary and secondary outcomes. The modified scale will be as follows:

- 8. Death;
- 7. Hospitalized, on invasive mechanical ventilation or ECMO;
- 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
- 5. Hospitalized, requiring supplemental oxygen;
- 4. Hospitalized, not requiring supplemental oxygen- requiring ongoing medical care (COVID-19 related or otherwise;
- 3. Not hospitalized, limitation on activities;
- 2. Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care; or Not hospitalized, no limitations on activities.

That is, category 1 and 3 of the original scale will be combined into the lowest category.

NEWS has demonstrated an ability to discriminate subjects at risk of poor outcomes. This score is based on 7 clinical parameters (see Section 8.1.2.3 in Appendix B of the study protocol). This should be evaluated at the first assessment of a given study day and prior to administration of study product. The 7 parameters can be obtained from the hospital chart using the last measurement prior to the time of assessment and a numeric score given for each parameter (e.g., a RR of 9 is one point, oxygen saturation of 92 is two points). This is recorded for the day obtained. i.e., on Day N, the Day N score is obtained and recorded as the Day N score.

Oxygenation, Non-invasive ventilation/high flow oxygen, Invasive Mechanical Ventilation / extracorporeal membrane oxygenation (ECMO), hospitalization and mortality will be assessed using results of the 8-point ordinal scale and post discharge eCRF questions.

Safety will be assessed by the following:

- Cumulative incidence of serious adverse events (SAEs) through 28 days of follow-up.
- Cumulative incidence of Grade 3 and 4 AEs.
- Discontinuation or temporary suspension of study product administration (for any reason)

• Changes in white cell count, absolute neutrophil count, hemoglobin, platelets, creatinine, glucose, total bilirubin, ALT, AST, and INR, d-dimer, C-reactive protein over time.

Clinical labs will be drawn on Days 1, 3, 5, 8, 11 and on Day 15 and 29 if the subject is able to return to the clinic or is still hospitalized.

Virologic efficacy is an exploratory endpoint and will be assessed by the following:

- Qualitative and quantitative PCR for SARS-CoV-2 in OP swab on Days 1; 3, 5, 8, 11 (while hospitalized); and Day 15 and 29 (if able to return to clinic or still hospitalized).
- Qualitative and quantitative PCR for SARS-CoV-2 in blood on Days 1; 3, 5, 8, 11 (while hospitalized).

To assess the impact of baricitinib on serum cytokine levels, blood samples will be assessed using a multiplex assay that is less sensitive to variability in sample integrity due to sample processing limitations during the pandemic. Cytokines to be tested may include (but not be limited to) IL-2, IL-19, IL-4, IL-10, IL-8, G-CSF, GM-CSF, MCP-1, MIP1 $\alpha$ , IL-7, IL-13, IL-31, IL-15, IL-6, IFN $\alpha$ , IFN $\gamma$  and TNF $\alpha$ . The list of cytokines tested is subject to change as new information about the pro-inflammatory state of COVID-19 is known. Given the challenges of obtaining samples and evolving knowledge about COVID-19, these will be considered exploratory endpoints. The description of the final methodology utilized, and the assay performance characteristics will be included in the final study report.

The schedule of study procedures is provided in Section 1.2 of Appendix B of the study protocol.

#### 5. SAMPLE SIZE CONSIDERATIONS

#### Sample Size for Primary Analysis

The log-rank test will be used to compare treatment arms with respect to time to recovery. For the log-rank test, the two key determinants of power are the total number of events (i.e., recoveries) E and the treatment-to-control ratio of the rate of recovery. The number of events required for power  $1 - \beta$  to detect a recovery rate ratio of  $\theta$  using a two-tailed test at alpha=0.05 is approximately

$$E = \frac{4(1.96 + z_{\beta})^{2}}{\{\ln(\theta)\}^{2}},$$

where  $z_{\beta}$  is the 100(1 –  $\beta$ )th percentile of the standard normal distribution.

The force of recovery (sometimes loosely referred to as the "recovery ratio") is the analogue of the hazard ratio and the term "recovery rate ratio" is the analogue of the hazard ratio in this setting. A recovery rate ratio of 1.31 was reported in Cao, Wang, Wen et al. (2020) for a lopinavir/ritonavir trial that used time to improvement by 2 categories as primary endpoint. A preliminary review of data from ACTT-1 demonstrated a recovery rate ratio 1.312. It is unlikely the second component of treatment will have a similar effect size. Therefore, a recovery ratio of 1.25 is assumed for this trial. A total of 723 recoveries are needed for a recovery ratio of 1.25 with 85% power. The study will accrue until approximately 723 recoveries have been achieved. The date of study closure will be estimated based on enrollment rate and recovery/enrollment percentages. If approximately 70% of participants recover, the total sample size will be 1032.

See Section 9.2 of Appendix B of the study protocol for discussions on the sample size calculations for the key secondary outcome.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

This is a double-blind, placebo controlled randomized trial with a two-sided type I error rate of 0.05. Secondary hypotheses have been ordered according to relative importance. These will be described according to the appropriate summary statistics, e.g.

- Percentages/proportions/odds ratios for categorical data. For tabular summaries of percentages/proportions, the denominator (e.g. number of subjects with non-missing data) will be displayed.
- Means, median, and range for continuous data, median for time-to-event data.

Confidence intervals will be generated; for the primary analysis, the confidence level will take into account the group-sequential design of the trial (see Section 6.6 and Section 8.1) whereas 95% confidence intervals will be generated for secondary and exploratory outcomes. For hazard ratio and odds ratio estimates, Wald confidence intervals will be used. For other efficacy outcomes, Wilson or Score confidence intervals will be used. For safety outcomes, exact (e.g. Clopper-Pearson) confidence intervals will be used.

When calculating treatment effects (e.g. differences, hazard ratios, odds ratios) and when using treatment arm as a covariate in regression modeling, the remdesivir+placebo arm will be used as the reference group. For regression modeling that uses strata variables defined in Section 6.4, the first stratum listed for each variable in that section will be used as the reference group.

For the final time-to-event analyses, the following SAS pseudocode will be used to perform stratified analyses to generate stratum-specific median time to event estimates and confidence intervals, stratum-specific Kaplan-Meier curves, and to perform the log-rank test. For any unstratified analyses, code can be used after the removal of the strata ...; line.

```
proc lifetest data=dataset plots=(s);
   time TimeVariable * CensorVariable(1);
   strata StrataVariable;
   test TreatmentVariable;
run;
```

Note that the interim efficacy analyses will be performed using R. For all interim and final analyses, the software used will calculate the log rank statistic using the formula in Section 8.1.1.

To perform a stratified Cox proportional hazards model for the final analysis and generate the treatment arm hazard ratio along with its confidence interval, the following pseudocode will be used. For any unstratified analyses, code can be used after the removal of the strata ...; line and strata variable in the class statement.

```
proc phreg data=dataset;
   class StrataVariable(ref=StrataLabel)
TreatmentVariable(ref=RemdesivirLabel);
   model TimeVariable * CensorVariable(1) = TreatmentVariable;
   strata StrataVariable;
   hazardratio TreatmentVariable / diff=ref cl=Wald;
   ods output HazardRatios = HRest;
run;
```

The following SAS pseudocode will be used to perform the final proportional odds model with treatment arm and disease severity as covariates and to generate the treatment odds ratio, p-value, and predicted probabilities of the ordinal scale levels by treatment arm and disease severity:

# **6.2.** Timing of Analyses

# **6.2.1.** Early Sample Size Reassessment

A blinded estimate of the proportion of recoveries will be computed during the trial to evaluate whether the total sample size will provide the number of recoveries.

# 6.2.2. Interim analyses

A DSMB will monitor ongoing results to ensure patient well-being and safety as well as study integrity. The DSMB will be asked to recommend early termination or modification only when there is clear and substantial evidence of a treatment difference. More details about the interim analyses are described in Section 6.6.1 and Section 6.6.2 below as well as a separate guidance document for the DSMB. The summaries to be generated for the interim analysis are provided in the separate DSMB shell report.

#### **6.2.3.** Final Analyses

The final analyses of all outcomes and planned summaries/listings will be performed on the final full locked database and provided in the final report.

# 6.3. Analysis Populations

Summaries and analysis of safety data will be presented for the As Treated Population. Summaries and analysis of efficacy data will be presented for the intent-to-treat (ITT) population and As Treated population.

#### 6.3.1. Intention-to-Treat (ITT) and As Treated Populations

The intent-to-treat (ITT) population includes all subjects who were randomized. For ITT analyses, subjects will be classified by their randomized treatment assignment and randomized disease severity stratum.

The As Treated population includes all randomized subjects who received the baricitinib/placebo study product, even if only one tablet was administered.

For As Treated analyses of efficacy outcomes, subjects will be classified by their actual treatment assignment and randomized disease severity stratum. Note that if no subjects are

administered the incorrect treatment, the As Treated efficacy analysis will not be performed as they will be identical to the ITT analyses.

For As Treated analyses of safety outcomes, concomitant medications, and medical history, subjects will be classified by their actual treatment assignment and actual disease severity stratum.

Note that per Section 6.4, subgroup analyses of outcomes will classify subjects by randomized (for safety outcomes) and actual (for efficacy outcomes) severity strata.

# 6.4. Covariates and Subgroups

Subgroup analyses for the main efficacy outcomes (i.e. the primary and key secondary analyses) will evaluate the treatment effect across the following subgroups:

- Geographic region:
  - o US sites: Non-US sites
  - o North American sites; Asian sites; European sites
- Duration of symptoms prior to enrollment
  - Quartiles
  - $\circ$  <= 10 days; > 10 days
  - <= Median; > Median
- Race (White; Black/African American; Asian; Other)
- Comorbidities
  - o None; Any
  - o None, One, Two or more
  - o Obese; Non-Obese
- Age (<40; 40-64; 65 and older),
- Sex (Female; Male),
- Severity of disease
  - o Randomization stratification: Moderate (ordinal 4/5); Severe (ordinal 6/7).
  - Actual disease severity at baseline: Moderate (ordinal 4/5); Severe (ordinal 6/7)
     Note these analyses will only be performed if at least one subject is erroneously randomized into the incorrect disease severity stratum.
  - o Baseline ordinal scale category: 4; 5; 6; 7

Additionally, main analyses of all secondary efficacy outcomes will evaluate the treatment effect across the following subgroups:

- Duration of symptoms prior to enrollment (<= Median; > Median)
- Severity of disease

- o Randomization stratification: Moderate (ordinal 4/5); Severe (ordinal 6/7).
- Actual disease severity at baseline: Moderate (ordinal 4/5); Severe (ordinal 6/7)
   Note these analyses will only be performed if at least one subject is erroneously randomized into the incorrect disease severity stratum.
- o Baseline ordinal scale category: 4; 5; 6; 7

There will also be a sensitivity analysis of the primary, key secondary, and mortality outcomes to evaluate the effect of concomitant therapy including experimental treatment and off-label use of marketed medications that are intended as treatment for COVID-19 and are given to patient prior to and during the study. A blinded review of the concomitant medication data will be performed by the medical monitor to identify medications that fall into any of the following categories of "Medications of Interest":

- Antivirals
  - Protease inhibitors
  - o Polymerase inhibitors
- Potential Treatments for COVID-19
  - o Hydroxychloroquine/Chloroquine
  - o Other
- Corticosteroids
- Other anti-inflammatory drugs
  - Monoclonal Antibodies Targeting Cytokines
  - Other Biologic Therapies

Summaries of subjects who report use of the categories and subcategories of therapies/treatments will be provided. Note that after the blinded review of the medications, additional categories/sub-categories may be defined and/or categories/sub-categories may be combined.

In addition, the sensitivity analyses will consider the following categories (individually):

- Any Medication of Interest
- Hydroxychloroquine/Chloroquine
- Corticosteroids
- Other Anti-Inflammatory Drugs

For the recovery analyses, if a subject recovered prior to use of any of the medications/therapies, then the subject will still be counted as a recovery in the sensitivity analysis. For the analysis of the key secondary outcome, if a subject reports use of any of the medications/therapies prior to their Day 15 assessment, then the subject's last clinical status score prior to medication/therapy use will be used as their Day 15 outcome. For the mortality analyses, subjects will be censored at the time of medication/therapy initiation.

In addition, the effect of treatment on the primary and key secondary efficacy outcomes will be explored via regression modeling controlling for age, duration of symptoms prior to enrollment, baseline d-dimer, and baseline CRP values as continuous covariates.

# 6.5. Missing Data

All attempts will be made to collect all data per protocol. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses may be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

For time to event outcomes, subjects who are lost to follow-up or terminate the study prior to Day 29 and prior to observing/experiencing the event will be censored at the time of their last observed assessment. Subjects who die prior to observing/experiencing the event will be censored at Day 29.

For the analysis of the key secondary outcome, subjects who are discharged but are subsequently re-admitted prior to Day 15 without a reported clinical score, their clinical score will be imputed at 7, which is the highest value for a hospitalized subject.

For the analyses of the secondary outcomes that involve clinical score (i.e. the key secondary outcome and time to improvement), if a subject is discharged from the hospital without a previously or concurrently reported clinical score of 1 or 2, then their clinical score at the time of discharge will be imputed as 2, which is the highest value for a non-hospitalized subject. If a subject terminates early from the study while they are hospitalized or completes the study while still hospitalized, the last observed clinical score assessment will be used as their final assessment.

For the modified version of the ordinal score described in Section 4.3, if a subject is discharged from the hospital without a previously or concurrently reported clinical score of 2 or 3, then their clinical score at the time of discharge will be imputed as 3, which is the highest value for a non-hospitalized subject.

For the analyses of the secondary outcomes described in Section 3.3, the following imputation rules will be used for subjects who are lost to follow-up, terminate early from the study, or do not have further outcome data available after discharge for any reason:

- Days of Non-invasive ventilation/high-flow oxygen:
  - o If the subject's clinical status scale is 6 at the last observed assessment, then the subject will be considered to be on non-invasive ventilation/high-flow oxygen through Day 29. The endpoint will be total days when assessments are available plus all imputed days following the last observed assessment.
  - o If the subject is <u>not</u> on non-invasive ventilation/high-flow oxygen at the last observed assessment, then the subject will be considered to <u>not</u> be on non-invasive ventilation/high-flow oxygen for the remainder of follow-up. Thus, no additional imputed days will be added to the number of days recorded on available assessments.

#### • Days of ventilation/ECMO:

- o If the subject's clinical status scale is 7 at the last observed assessment, then the subject will be considered to be on ventilation/ECMO through Day 29. The endpoint will be total days when assessments are available plus all imputed days following the last observed assessment.
- If the subject is not on ventilation/ECMO at the last observed assessment, then the subject will be considered to not be on ventilation/ECMO through Day 29. Thus, no additional imputed days will be added to the number of days recorded on available assessments.

# • Days of Oxygen:

- o If the subject's clinical status score is 5, 6, or 7 at the last observed assessment, then the subject will be considered to be on oxygen through Day 29. The endpoint will be total days when assessments are available plus all imputed days following the last observed assessment.
- o If the subject is not on oxygen at the last observed assessment, then the subject will be considered to not be on oxygen through Day 29. Thus, no additional imputed days will be added to the number of days recorded on available assessments.

# • Days of Hospitalization

o If the subject is discharged and no further hospitalization data are available, then the subject will be assumed to not have been readmitted. Thus, no additional imputed days will be added to the number of days recorded on available assessments. If a subject dies while hospitalized, the number of days of hospitalization will be imputed as 28 days.

# 6.6. Interim Analyses and Data Monitoring

#### 6.6.1. Interim Safety Analyses

Interim safety data will be available electronically in real time. No formal interim safety analyses are planned.

#### 6.6.2. Interim Efficacy Review

An interim efficacy analysis will be conducted after approximately 33% of total information has been reached. The information fraction at an interim analysis will be computed as t = r/723 where r is the number of recoveries by the time of the data freeze date for the interim analysis. The Lan-DeMets spending function analog of the O'Brien-Fleming boundary will be used to monitor the primary endpoint using an overall two-sided type-I error rate of 0.05. Specifically, two one sided boundaries are constructed at level 0.025 using the spending function

$$\alpha^*(t) = 2[1 - \Phi\{2.241/t^{\frac{1}{2}}\}],$$

where  $\Phi$  is the standard normal distribution function. Lan-DeMets software from the University of Wisconsin, now available in the R package 'ldbounds', will be used to calculate boundaries.

Conditional power will be presented as an additional guide to the DSMB. Conditional power allows computation of the probability of obtaining a statistically significant result by the end of the trial given the data accumulated thus far, incorporating and assuming a hypothesized treatment effect (e.g., the treatment effect assumed for sample size determination) thereafter. If conditional power is less than 20% under the original trial assumptions, consideration should be given to stopping the trial.

The unblinded statistical team will prepare these closed session reports for DSMB review and recommendations. Analyses will be presented with blinded codes for treatment arms to protect against the possibility that the DSMB report may fall into the wrong hands. A DSMB Charter will further describe procedures and membership. An additional document on statistical issues related to monitoring may be provided to the DSMB prior to interim analyses.

#### 6.7. Multicenter Studies

Data will be pooled across all clinical sites. Secondary analyses of the primary outcome will account for site via stratification by geographic region as noted in Section 6.4.

A sensitivity analysis of the primary outcome will be performed to assess the impact of individual sites on the observed treatment effect. Letting M be the total number of sites, the primary analysis will be repeated by excluding a single clinical site and performing the analyses on the remaining M-1 sites. This process will be repeated so that estimates are generated for each of the M-1 subset datasets. Presentations from these analyses are described in Section 8.1.2.

# 6.8. Multiple Comparisons/Multiplicity

There is only one primary outcome measure. The study utilizes a group-sequential design to control the overall type I error rate while allowing for formal interim analyses of the primary outcome measure (as described in Section 6.6 and Section 8.1). There is no planned adjustment for multiple comparisons in any secondary or exploratory analyses.

#### 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

A summary of the reasons that subjects were screened but not enrolled will be tabulated (Table 1).

The composition of analysis populations, including reasons for subject exclusion will be summarized by treatment group and disease severity (Table 2). A subject listing of analysis population eligibilities will be generated (Listing 1).

The disposition of subjects will be tabulated by treatment group and disease severity (Table 3). Study milestones included in the table will include, but not limited to: the total number of subjects that were randomized, completed expected blood draws, completed Study Day 15 visit, completed Study Day 22 visit, and completed Study Day 29 visit. For the calculation of percentages, subjects who die will not be included in the denominators for visits/assessments beyond their death.

Treatment compliance will be summarized by treatment group (Table 4). Summaries of prior Remdesivir treatment by treatment group will also be provided (Table 5 and Table 6)

A flowchart showing the disposition of study subjects, adapted from the Consort Statement [4] will be generated (Figure 1). This figure will present the number of subjects screened, randomized, lost to follow-up, and analyzed, by treatment group and disease severity.

A listing of subjects who discontinued dosing or terminated study follow-up and the reason will be generated (Listing 2).

#### 7.2. Protocol Deviations

Subject-specific protocol deviations will be summarized by the reason for the deviation, the deviation category, treatment group, disease severity and (separately) geographic region for all subjects (Table 7 and Table 8). Supplementary protocol deviation summaries will also be generated (e.g. major deviations, non-subject specific deviations). All subject-specific protocol deviations and non-subject specific protocol deviations will be included in listings (Listing 3 and Listing 4).

#### 8. EFFICACY EVALUATION

# 8.1. Primary Efficacy Analysis

# 8.1.1. Primary Analyses

The primary analysis uses the stratified log rank test to compare treatment to control through Day 29 with respect to time to recovery, as defined in Section 3.3. Stratification is based on moderate versus severe disease at baseline. As noted in Section 3.3, all deaths within 29 days will be considered censored at Day 29 with respect to time to recovery. Conceptually, a death corresponds to an infinite time to recovery, but censoring at any time greater than or equal to Day 29 gives the same answer as censoring at Day 29; both correspond to giving deaths the worst rank.

Let MM and S denote the Moderate and Severe subgroups, respectively. The z-score associated with the stratified log rank test is

$$Z = \frac{\sum_{MM} (O_i - E_i) + \sum_{S} (O_i - E_i)}{\sqrt{\sum_{MM} V_i + \sum_{S} V_i}}.$$

The sums are over recovery times  $t_i$  in the moderate and severe subgroups,  $O_i$  is the number of treatment arm participants recovering at time  $t_i$ , and  $E_i$  and  $V_i$  are the null expected value and variance of the number of treatment recoveries calculated using the hypergeometric distribution. Specifically, if  $n_{Ti}$  and  $n_{Ci}$  denote the numbers of patients 'at risk' in the two arms in a given stratum at  $t_i$ , and  $r_i$  is the total number of recoveries at  $t_i$ , then  $E_i = r_i n_{Ti} / (n_{Ti} + n_{Ci})$  and  $V_i = r_i (n_i - r_i) n_{Ti} n_{Ci} / [n_i^2 (n_i - 1)]$ , where  $n_i = n_{Ti} + n_{Ci}$ . The  $O_i$ ,  $E_i$ , and  $V_i$  are computed separately within the moderate and severe strata.

As noted in Section 6.6.2, to maintain an overall two-sided type-I error rate of 0.05, the Lan-DeMets spending function analog of the O'Brien-Fleming boundary will be used to derive the cumulative error spending and boundaries for the interim analysis.

For the final analysis, the log rank test will be performed using the pseudocode provided in Section 6.1. The following pseudocode can be used to compute the bounds for the final analyses and compare to the calculated log-rank statistic. The Boundaries dataset will contain the updated boundaries calculated from the interim analyses using the actual information levels observed at the interim analysis.

ods output Test=FinalResults ParameterEstimates = LogHRest;
run;

If the trial is stopped at the interim analysis, then to derive the p-value, hazard ratio estimate, and confidence interval for the early and final analysis sets, stage-wise ordering of the sample space will be used [5]. The resulting p-value, median unbiased estimate, and confidence interval will be presented in the final report. If the trial is not stopped early, then the fixed sample estimates of the statistics using an alpha level of 5% will be computed and reported for the final analysis. The SAS pseudocode above provides estimates for the log hazard ratio and so the estimates will be exponentiated and reported.

The primary analysis will be performed in the ITT analysis population. The treatment hazard ratio estimate and confidence interval and p-value from the stratified log rank test will be presented (Table 15). The median time to event and 95% confidence interval will be summarized by treatment arm and disease severity. In addition, stratum-specific estimates of the treatment hazard ratio from Cox models run within each of the disease severity strata will be presented. Kaplan-Meier curves for each treatment arm will be presented, supplemented with the hazard ratio estimate, p-value, and the number of subjects at risk in each arm and severity stratum at Days 1, 3, 5, 7, 11, 15, 22, and 29 (Figure 2).

Subject listings of the ordinal scale results by day will be generated (Listing 5).

# 8.1.2. Supplemental and Sensitivity Analyses

For all supplemental and sensitivity analyses of the primary outcome, p-values may or may not be reported, and 95% confidence levels will be used for confidence interval estimates.

The primary analysis will be repeated in the As Treated analysis population where subjects who are not treated will be censored at enrollment. The tabular and graphical summaries described in the previous section will be replicated for this As Treated analysis.

Sensitivity analyses will be performed using Cox proportional hazards models to estimate the hazard ratio. First, an ITT analysis will be performed in which subjects who die prior to recovering are treated as experiencing a competing risk in the Fine-Gray proportional hazards regression model. Second, a Cox model will be fit with binary indicators for treatment group and disease severity Moderate vs. Severe [separate models for randomized stratum and actual stratum]) as well as a treatment \* disease severity interaction term. The models will be fit to the ITT analysis population. The treatment group hazard ratios and CIs will be reported for both sets of models and the interaction term p-value will be reported for the interaction models. As requested by the DSMB, a restricted mean survival time analysis will be performed as an exploratory analysis. The restricted mean recovery time estimates will be provided for each treatment group and randomized disease severity stratum as well as the difference in restricted mean recovery time between treatment groups within each of the severity strata (Table 18). Time to recovery will also be explored within prior Remdesivir treatment subgroups (Any Treatment vs. No Treatment) (Table 19).

The primary analysis will also be repeated using the other subgroups defined in Section 6.4 in place of disease severity. Each subgroup will be considered separately and the tabular and graphical summaries described in the previous section will be replicated for each subgroup. The tabular summary will also include results from an analysis of time to recovery controlling for age

and duration of symptoms as continuous covariates and baseline d-dimer and CRP values as continuous covariates. A forest plot will be generated to display the overall treatment hazard ratio estimate and CI from each of the within-stratum analyses (Table 20 and Table 21). These analyses will be performed in the ITT and As Treated populations.

In addition, a forest plot will be generated for the "leave one out" sensitivity analyses described in Section 6.7; hazard ratio estimates and CIs will be provided for each subgroup that leaves a single site out.

An additional sensitivity analysis will evaluate the effect of recoveries that were not sustained as indicated in Section 3.3.2.

As noted in Section 6.4, analyses that take into account concomitant medication will be performed. The primary analysis will be repeated, where subjects who take prohibited medications will be treated as treatment failures and will be censored at the time of medication use.

Two corroborative summaries will also be generated. A summary of the number and percentage of subjects in each treatment group who recovered (and are alive), did not recover (and are alive), and died by Day 29 will be summarized. The summary will also include the numbers and percentages, grouping deaths and non-recoveries together (Table 24). The summaries will also be provided by the duration of symptoms categorizations specified in Section 6.4.

Other censoring techniques and additional analyses of the primary outcome may be performed.

# 8.2. Secondary Efficacy Analyses

This section describes the planned analyses for the secondary efficacy outcome measures. Where applicable, refer to Section 6.1 for SAS pseudocode. Analyses of mortality will be described in Section 9.4.

Analyses of the key secondary outcome measure will be explored in the specified subgroups described in Section 6.4. Analyses of the other secondary outcome measures will be performed by treatment arm only and repeated for specified subgroups described in Section 6.4 and Section 6.7 via stratified analyses. As with the analyses described in Section 8.1.2, tabular summaries will follow the structure of the main tabular summaries planned for each outcome with the modification that stratified estimates will be provided in separate rows. Forest plots will display confidence intervals of outcomes/estimates across subgroups, where applicable.

All secondary efficacy analyses will be performed in the ITT population. As Treated analyses will be explored to investigate consistency of results compared to the ITT analyses.

# 8.2.1. Ordinal Scale Outcomes (Key Secondary Outcome Measure)

For the analysis of the key secondary outcome measure, the distribution of the 8-point ordinal clinical status scale with 8 categories at Study Visit Day 15 (not necessarily actual study day 15), the outcome will be analyzed using a proportional odds model with treatment arm and disease severity as covariates. The treatment odds ratio estimated from the model will be presented along with the p-value (Table 25). The Study Visit Day 15 clinical status score will be depicted graphically using shifted bar plots; the outcomes will be presented by baseline ordinal score and treatment group (Figure 13). In addition to the subgroup analyses, the main analysis will be

repeated including a treatment \* disease severity interaction term, where the interaction term p-value will be reported for the interaction model.

Multiple supplemental analysis of this key secondary outcome will be performed. Time to improvement by at least one category in the clinical status 8-point scale (see Section 3.3). The log rank test will be performed using a Cox proportional hazards model to test whether the curves differ between treatment arms. The median time to event and CI in each treatment group will be summarized along with the treatment hazard ratio estimate and log rank p-value (Table 27). Differences in time-to-event endpoints by treatment arm will be summarized with Kaplan-Meier curves (Figure 16). Number at risk, hazard ratio and log rank p-values will be presented on the figures. The analyses (and tabular and graphical summaries) will be repeated using the outcome of time to improvement in two categories of the ordinal scale defined in Section 3.3. In addition, a subgroup analysis time to improvement among subjects enrolled with a clinical score of 7 will be performed using the retreatment censoring plan.

The above analyses will be repeated with the modification to the ordinal scale described in Section 4.3 (Table 28).

The number and proportion of subjects along with 95% confidence intervals by category of clinical status will be presented by treatment arm at Study Visit (not necessarily actual) Days 1, 3, 5, 8, 11, 15 and 29 (Table 33). Change from baseline will also be summarized at Days 3, 5, 7, 11, 15, 22, and 29 (Table 35). A figure will present stacked bar charts by day with side by side bars for each treatment arm (Figure 25). Histograms will be generated to display the ordinal scale value distributions over time in each treatment group (Figure 26).

#### *8.2.2.* NEWS

The median time to discharge or to a NEWS of  $\leq 2$  and CI will be summarized by treatment group (Table 37). The hazard ratio and log rank p-values will be provided with the summaries. Differences in time-to-event endpoints by treatment arm will be summarized with Kaplan-Meier curves. Number at risk, hazard ratio and log rank p-values will be included on the figures (Figure 27).

The mean, standard deviation (SD), median, minimum, and maximum NEWS at Baseline and Study Visit (not necessarily actual) Days 3, 5, 8, 11, 15 and 29 will be presented by treatment arm as well as change from baseline at each post-Day 1 visit (Table 40). A figure with mean and SD over time will also be presented by treatment arm (Figure 32).

Subject listings of NEWS responses (overall and individual components) by day will be generated (Listing 6).

#### 8.2.3. Days of Oxygenation

Duration of oxygenation days will be summarized in a table using medians and quartiles by treatment arm (Table 42). This will only include subjects in category 5, 6, or 7 at randomization. Analyses will be performed in the ITT and As Treated populations. Bee swarm plots of oxygen days by treatment arm will be generated, where subjects whose days are imputed to the maximum of 28 days due to death are grouped separately from subjects who do not die (Figure 33).

# 8.2.4. Incidence of New Oxygen use

The incidence and duration of new oxygen use will be analyzed by treatment arm. This will only include subjects in category 4 at randomization. New use will be identified by a post-enrollment score of at least 5; the number of subjects reporting new use and the incidence rate (and CI) will be reported.

#### 8.2.5. Days of Non-Invasive Ventilation/High-Flow Oxygen

Duration of non-invasive ventilation/high flow oxygen days will be summarized in a table using medians and quartiles by treatment arm. This will only include subjects in category 6 at randomization. Analyses will be performed in the ITT and As Treated populations. Bee swarm plots of non-invasive ventilation/high flow oxygen days by treatment arm will be generated, where subjects whose days are imputed to the maximum of 28 days due to death are grouped separately from subjects who do not die.

# 8.2.6. Incidence of New Non-Invasive Ventilation/High-Flow Oxygen

The incidence and duration of new Non-Invasive Ventilation/High-Flow Oxygen use will be analyzed by treatment arm. This will only include subjects in category 4 or 5 at randomization. New use will be identified by a post-enrollment score of 6. The number of subjects reporting new use and the incidence rate (and CI) will be reported.

# 8.2.7. Days of Invasive Mechanical Ventilation/ECMO

Duration of invasive Mechanical Ventilation/ECMO days will be summarized in a table using medians and quartiles by treatment arm. This will only include subjects in category 7 at randomization. Analyses will be performed in the ITT and As Treated populations. Bee swarm plots of invasive Mechanical Ventilation/ECMO days, and days hospitalized by treatment arm will be generated, where subjects whose days are imputed to the maximum of 28 days due to death are grouped separately from subjects who do not die.

# 8.2.8. Incidence of New Invasive Mechanical Ventilation/ECMO

The incidence and duration of new Invasive Mechanical Ventilation/ECMO use will be analyzed by treatment arm. This will only include subjects in category 4, 5, or 6 at randomization. New use will be identified by a post-enrollment score of 7. The number of subjects reporting new use and the incidence rate (and CI) will be reported.

#### 8.2.9. Days of Hospitalization

Duration of hospitalization days will be summarized in a table using medians and quartiles by treatment arm. Incidence of readmittance will also be summarized (Table 48). Analyses will be performed in the ITT and As Treated population. Bee swarm plots of days hospitalized by treatment arm will be generated, where subjects whose days are imputed to the maximum of 28 days due to death are grouped separately from subjects who do not die.

# 8.3. Exploratory Efficacy Analyses

Analyses of exploratory outcome measures are not covered in this SAP.

# 9. SAFETY EVALUATION

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, height, weight, BMI, ethnicity, and race will be presented by treatment group as well as geographic region, comorbidities, duration of symptoms prior to enrollment, and disease severity (Table 50 and Table 51). Ethnicity will be categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option.

Individual subject listings will be presented for all demographics and baseline characteristics (Listing 7).

#### 9.1.1. Prior and Concurrent Medical Conditions

Focused medical history is obtained at the screening visit that includes the following:

- History of chronic medical conditions related to inclusion and exclusion criteria
- Review medications and therapies for this current illness.

Medical history is limited to the following conditions: asthma, cancer, cardiac valvular disease, chronic kidney disease, chronic liver disease, chronic oxygen requirement, chronic respiratory disease, coagulopathy, congestive heart failure, coronary artery disease, current nicotine consumption, diabetes I and II, hypertension, immune deficiency, obesity, and risk for deep vein thrombosis (DVT) or pulmonary embolism (PE). All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 23.0 or higher. Summaries of subjects' pre-existing medical conditions will be presented by treatment group (Table 52).

Individual subject listings will be presented for all medical conditions (Listing 8).

#### 9.1.2. Prior and Concomitant Medications

Medication history (concomitant medications) includes a review of all current medications and medications taken within 7 days prior to enrollment through approximately Day 15 or early termination (if Day 15), whichever occurs first.

Summaries of medications that were started prior to dosing and continued at the time of dosing or started after dosing while on study will be presented by WHO Drug Level 1 and 2 Codes, disease severity, and treatment group (Table 53). Summaries of overall use of prohibited medications/therapies listed in Section 6.4 that were started prior to dosing and continued at the time of dosing or started after dosing while on study as well as use by select study days will also be generated (Table 54 and Table 55).

Individual subject listings will be presented for all concomitant medications (Listing 9).

# **9.2.** Measurements of Treatment Compliance

Table 4 will provide summaries of key treatment compliance milestones/variables. In addition, the number of subjects with halted, slowed, or missed doses will be summarized by treatment arm (See Section 7).

Individual subject listings will be presented for all subjects who discontinued dosing (Listing 2). Individual subject listings will be presented for all subjects who missed, halted or slowed any doses (Listing 10).

#### 9.3. Adverse Events

For the calculation of incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the number of subjects in the Treated population. All adverse events reported will be included in the summaries and analyses.

An overall summary by treatment arm and disease severity of adverse events is presented that includes, but not limited to: subjects with at least one event, at least one related event, at least one SAE, at least one related SAE and at least one AE leading to early termination (Table 56 and Table 57).

Adverse events occurring in 5% of subjects (by MedDRA preferred term) in any treatment group will be presented (Table 58).

The proportion of subjects reporting at least one adverse event will be summarized by MedDRA system organ class and preferred term for each treatment arm, disease severity and overall. Denominators for percentages are the number of subjects in the Treated population.

The following summaries for adverse events will be presented by MedDRA system organ class, preferred term, disease severity and treatment group:

- Treatment-emergent renal adverse events by preferred term (Table 61);
- Treatment-emergent hepatic adverse events by preferred term (Table 62);
- Related adverse events by MedDRA system organ class and preferred term (Table 63);
- Subject listing of non-serious adverse events (Listing 11);
- Bar chart of non-serious related adverse events by severity and MedDRA system organ class (Figure 37);
- Bar chart of non-serious related adverse events by maximum severity and MedDRA system organ class (Figure 40);

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

Listings of death and other serious adverse events will be presented, including Subject ID, treatment group, Adverse Event Description, Number of Days Post Dose (Duration), Number of Days Post Dose the Event Became Serious, Reason Reported as an SAE, Severity, Relationship
to Treatment, Alternate Etiology if not Related, Action Taken with Study Treatment, Subject Discontinuation, Outcome, MedDRA SOC, and MedDRA PT (Listing 14 and Listing 16).

The number of subjects who die by Day 15 and Day 29 will be presented by treatment arm. The 14- and 28-day mortality rate, which will use Kaplan-Meier estimator, will be presented (Table 64).

Mortality through Day 15 and 29 will also be analyzed as a time to event endpoint (see Section 3.3). A table will present median time to event along with 95% confidence intervals overall for each treatment arm along with the hazard ratio estimate and log rank p-values (Table 66). Differences in time-to-event endpoints by treatment will be summarized with Kaplan-Meier curves (Figure 44). Analyses of mortality will be performed in the ITT and the Treated analysis populations. As a supplemental analysis, a Cox model will be fit with binary indicators for treatment group and disease severity as well as a treatment \* disease severity interaction term. The model will be fit in the ITT and Treated analysis populations. The treatment group hazard ratios and CIs and the interaction term p-value will be reported. Finally, the results of the sensitivity time-to event analysis described in Section 6.4 will be presented in a table; the same summaries as in Table 66 will be provided. As requested by the DSMB, a restricted mean survival time analysis of mortality will be performed as an exploratory analysis. The restricted mean mortality time estimates will be provided for each treatment group and randomized disease severity stratum as well as the difference in restricted mean recovery time between treatment groups within each of the severity strata (Table 72).

Rates of Grade 3 and 4 AE occurrence will be compared between treatment arms using Barnard's exact test and presented. Rates of SAE occurrence will also be compared between treatment arms using Barnard's exact test and presented. Further, the composite endpoint of the occurrence of death, SAE, or Grade 3 or 4 AE described in Section 3.3 will be analyzed as a time to event outcome. A table will present median time to event along with 95% confidence intervals overall for each treatment arm along with the hazard ratio estimate and log rank p-values (Table 73). Differences in time-to-event endpoints by treatment will be summarized with Kaplan-Meier curves.

A summary of the infections reported on the AE CRF will be summarized by treatment group and disease severity (Table 74). The anatomical location(s) of the infection and causative pathogen(s) determined by culture will be summarized. Infections considered to be opportunistic, as identified by the sponsor, will also be included in the summaries.

# 9.5. Pregnancies

For any subjects in the Treated population who become pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. Note that the CSR will not be delayed to wait for outcomes of any pregnancies; an addendum to the CSR would be provided in such a scenario. A set of listings of pregnancies and outcomes will be presented (Listing 14, Listing 15, Listing 16, Listing 17, and Listing 18).

# 9.6. Clinical Laboratory Evaluations

Clinical safety laboratory adverse events are collected Day 1, 3, 5, 8, 11 and Day 15 and 29 if able to return to clinic or still hospitalized. Parameters evaluated include white blood cell count, absolute neutrophil count, eGFR, platelet count, hemoglobin concentration, creatinine, glucose, total bilirubin, ALT, AST, INR, d-dimer, and CRP. Laboratory safety parameters will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, version 2.1 (July 2017).

The distribution of Grade 3 and 4 chemistry and hematology laboratory results by maximum severity, time point, disease severity and treatment group will be presented (Table 80). Treatment-emergent laboratory abnormalities will be summarized by parameter and grade (Table 83).

Descriptive statistics including mean, median, standard deviation, maximum, and minimum values and change from baseline by time point, for all and each chemistry and hematology laboratory parameter will be summarized by disease severity and treatment arm (Table 84). Changes in chemistry and hematology laboratory values will be presented in line graphs over time with mean and SD plotted by disease severity and treatment arm (Figure 53).

Listings will provide a complete listing of individual chemistry and hematology laboratory results with applicable reference ranges (Listing 19).

# 9.7. Vital Signs and Physical Evaluations

Vital sign measurements include pulse, systolic blood pressure, respiratory rate, SpO<sub>2</sub> and oral temperature. Vital signs were assessed as part of the NEW score (assessed daily while hospitalized and on Day 15) and will be listed in Listing 6.

Targeted Physical examinations are performed at Day 1 and are performed post-baseline only when needed to evaluate possible adverse events. At the screening visit, the targeted physical examination is focused on lung auscultation. Physical exam findings per subject will be detailed in a listing (Listing 20).

#### 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. Concomitant medication use will be presented in a subject listing (Listing 9). The use of concomitant medications during the study (regardless of whether the medications were started prior to enrollment or after enrollment) will be summarized by ATC1, ATC2 code, disease severity and treatment group for the Treated population (Table 53).

# 9.9. Other Safety Measures

No additional safety analyses are planned.

# 10. PHARMACOKINETICS

Not applicable.

# 11. IMMUNOGENICITY

Not applicable.

# 12. OTHER ANALYSES

Not applicable.

#### 13. REPORTING CONVENTIONS

P-values  $\ge 0.001$  and  $\le 0.999$  will be reported to 3 decimal places; p-values less than 0.0005 will be reported as "< 0.001" and p-values greater than 0.9995 will be reported as "> 0.999".

The mean, standard deviation, median, IQR, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data.

Proportions will be presented as 2 decimal places; values greater than zero but <0.005 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 0.5% will be presented as "<1"; values greater than 99.5% but less than 100% will be reported as >99.

Estimated parameters, not on the same scale as raw observations (e.g. hazard ratios and regression coefficients) will be reported to 3 significant figures.

# 14. TECHNICAL DETAILS

SAS version 9.4 or above, or R language and environment for statistical computing 3.6.1 or above, will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

The below summarizes the changes made to the SAP from version 2.0 to version 3.0:

In performing the final analyses of the ACTT-1 data, multiple tabular and graphical output required modifications from the shells provided in the ACTT-1 SAP to fixes errors, make clarifications, and provide additional supplementary information. After review of the analyses for ACTT-1, multiple ad-hoc analyses were also performed as requested by the sponsor, manufacturer, and FDA. In addition, exploratory analyses of the primary outcome were requested by the ACTT-2 DSMB. The modifications to the ACTT-1 shells as well as the additional analyses requested for ACTT-1 has been added to this version of the ACTT-2 SAP. The additional analyses are all supplemental exploratory analyses and were not driven by review of the ACTT-2 data but were added to provide consistent analyses and summaries across the individual ACTTs.

The additional summaries were added to the TFL appendices of this SAP; general updates were made to the corresponding text within the body of the document, however granular details of each new output were not necessarily added. Note that in adding the additional TFLs, a large number of the existing TFLs were renumbered to conform to eCTD guidelines.

#### Throughout the document:

- Typos and errors introduced via copying/pasting language from other sections were corrected.
- The Treated Population was renamed as the "As Treated Population".
- It was clarified that analyses that explore and/or incorporate readmittance will only consider readmittances for COVID-19 reasons.

#### Section **6.3.1**:

• The definitions of the analysis populations were clarified to explicitly denote when the randomized treatment assignment or disease severity stratum would be used versus the actual treatment group or disease severity. TFL shells were updated to explicitly state whether randomized or actual group/severity will be used.

#### Section 6.4:

• The process for identifying the medications of interest and the categories of medications were updated to match what was used for ACTT-1. Corresponding TFLs were updated accordingly.

## Appendices:

- Multiple TFLs were updated to fix omissions/errors and provide additional programming notes.
- The formatting of multiple TFLs was updated to provide better organized and/or more clear displays of the content.

#### Table 3:

• Included summaries and format was updated to match those used for the corresponding final ACTT-1 table.

#### Table 4:

- Replaced the term "Completed" with "Received" for infusion summaries throughout.
- Summaries of prior RDV treatment were added.

#### Table 5 and Table 6:

• Multiple additional protocol deviation tables were added to match those generated for ACTT-1.

#### Table 16 and Table 17:

• Ad-hoc Fine-Gray, Covariate-Adjusted, and Interaction Modeling analyses of time to recovery were added to match those performed for ACTT-1.

#### Table 18:

• Restricted Mean Survival Time analysis of time to recovery was added per request by the ACTT-2 DSMB.

#### Table 19:

• Ad-hoc analysis of time to recovery by prior RDV treatment was added.

#### Table 35 and Table 36:

• Summaries of clinical status score at individual time points was added to match those generated for ACTT-1.

#### Table 42, Table 43, Table 44, Table 45, Table 46, Table 47:

 Tables were updated to provide additional summaries which were provided in the ACTT-1 final analyses.

#### Table 51:

• IQR was added to match the addition to the corresponding table in ACTT-1.

#### Table 56 and Table 57:

• Additional key safety event categories were added to the table as was requested for ACTT-1. In addition, a table summarizing the risk difference of a subset of these events (difference between treatment groups) was added per request for ACTT-1.

#### Table 61, Table 62, Table 63:

• Additional summaries of adverse event data were added to match the additions to the ACTT-1 final analyses, including renal AEs, hepatic AEs, and related AEs.

#### Table 64, Table 65, Table 66, Table 67:

• Disease Severity was added to the tabular summaries.

#### Table 71:

• Restricted Mean Survival Time analysis of time to death was added per request by the ACTT-2 DSMB.

#### Table 75, Table 77, Table 79:

• Opportunistic infection summaries were added; shells were erroneously omitted from previous versions of the SAP.

#### Table 80, Table 81, Table 82, Table 83:

• A column for Grade 3 or 4 was added as the column was added to the corresponding ACTT-1 table. In addition, disease severity-specific summaries and summaries of treatment-emergent laboratory abnormalities were added, as similar summaries were generated for ACTT-1.

#### Table 85 and Table 86:

• Disease severity-specific summaries were added.

#### Figure 6, Figure 7, Figure 8, Figure 9:

• Figures displaying time to recovery Kaplan-Meier curves within subgroups defined by baseline ordinal score were added to match the figures generated for ACTT-1.

#### Figure 12:

• Forest plot of the hazard ratios of time to recovery by comorbidity was added to match the figure generated for ACTT-1.

#### Figure 17, Figure 18, Figure 19, Figure 20, Figure 21, Figure 22, Figure 23, Figure 24:

• Figures displaying time to improvement Kaplan-Meier curves within subgroups defined by baseline ordinal score were added to match the figures generated for ACTT-1.

#### Figure 28, Figure 29, Figure 30, Figure 31:

• Figures displaying time to discharge or NEWS <= 2 Kaplan-Meier curves within subgroups defined by baseline ordinal score were added to match the figures generated for ACTT-1.

#### Figure 44 and Figure 46:

• Figures displaying time to death Kaplan-Meier curves within subgroups defined by disease severity and baseline ordinal score were added to match the figures generated for ACTT-1.

#### Figure 47, Figure 48, Figure 49, Figure 50:

• Figure displaying time to death Kaplan-Meier curves within subgroups defined by disease severity was added.

#### The below summarizes the changes made to the SAP from version 1.0 to version 2.0:

#### Throughout the document:

• Typos and errors introduced via copying/pasting language from other sections were corrected.

#### Section 3.3.2:

Language was added to the definition of recovery to note that subjects who are
discharged to another hospital, hospice, or similar health care institution will not be
considered recovered.

#### Section 6.4:

• The Prohibited Medications that are being explored in sensitivity analyses were renamed "Medications of Interest". Corresponding tables and listings were updated accordingly.

#### Section 6.5:

• Language was added to the imputation rules for clinical scores to note that if a subject terminates early from the study while they are hospitalized or completes the study while still hospitalized without a reported clinical score on the day of discharge, the last observed clinical score assessment will be used as their final assessment.

#### Section 9.4:

• A supplemental analysis of the time to death outcome was added to explore the interaction between treatment and baseline disease severity with respect to the effect of treatment on the outcome.

#### Appendices:

• Multiple tables and listings were updated to fix omissions/errors and provide additional programming notes.

## 16. REFERENCES

- 1. Schoenfeld, D. 1981. The asymptotic properties of nonparametric tests for comparing survival distributions. Biometrika. 68 (1): 316–319.
- 2. Cao, Wang, Wen et al. 2020. A trial of lopinavir—ritonavir in adults hospitalized with severe covid-19. New DOI: 10.1056/NEJMoa2001282.
- 3. Whitehead, J. 1993. Sample size calculations for ordered categorical data. Statistics in Medicine 12, 2257-2271.
- 4. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.
- 5. Jennison C., Turnbull B.W. 2000. Group sequential methods with applications to clinical trials. Chapman & Hall, Boca Raton.

# 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

The formatting of the final version of a table, figure, or listing may differ from what is presented in the shell or the presentation of the results may be changed, however the key content will remain unchanged. Additional summaries/data points may be included in the final version of a table, figure, or listing, as well. Additional tables, figures, and listings may be generated to supplement the planned output.

# APPENDIX 1. TABLE MOCK-UPS

# LIST OF TABLES

| Table 1: | Ineligibility Summary of Screen Failures | 55 |
|---|---|---|
| Table 2: | Analysis Population Eligibilities by Treatment Group and Randomized Disease Severity | 56 |
| Table 3: | Subject Disposition by Treatment Group and Randomized Disease Severity – ITT Population | 57 |
| Table 4: | Treatment Compliance by Treatment Group | 58 |
| Table 5: | Subjects Reporting Prior Remdesivir Treatment by Randomized Disease<br>Severity and Treatment Group – ITT Population | 60 |
| Table 6: | Subjects Reporting Prior Remdesivir Treatment by Actual Disease Severity and Treatment Group – As Treated Population | 60 |
| Table 7: | Distribution of Subject Specific Protocol Deviations by Category, Type, Treatment Group, and Randomized Disease Severity | 61 |
| Table 8: | Distribution of Subject Specific Protocol Deviations by Category, Type, and Geographic Region | 63 |
| Table 9: | Distribution of Major Subject Specific Protocol Deviations by Category, Type, Treatment Group, and Randomized Disease Severity | 63 |
| Table 10: | Distribution of Major Subject Specific Protocol Deviations by Category, Type, and Geographic Region | 63 |
| Table 11: | Distribution of Non-Subject Specific Protocol Deviations by Category and Type | 63 |
| Table 12: | Distribution of Non-Subject Specific Protocol Deviations by Category, Type, and Geographic Region | 63 |
| Table 13: | Distribution of Major Non-Subject Specific Protocol Deviations by Category and Type | 63 |
| Table 14: | Distribution of Major Non-Subject Specific Protocol Deviations by Category, Type, and Geographic Region | 63 |
| Table 15: | Time to Recovery by Treatment Group and Randomized Disease Severity | 64 |
| Table 16: | Time to Recovery by Treatment Group and Randomized Disease Severity: Fine-Gray, Covariate-Adjusted, and Interaction Modeling | 64 |
| Table 17: | Time to Recovery by Treatment Group and Baseline Ordinal Score: Fine-Gray and Interaction Modeling | 64 |
| Table 18: | Time to Recovery by Treatment Group and Disease Severity: Restricted Mean Survival Time Analysis – ITT Population | 65 |

| Table 19: | Time to Recovery by Treatment Group within Prior RDV Treatment Subgroups | 65 |
|---|---|---|
| Table 20: | Time to Recovery by Treatment Group within Subgroups – ITT Population | 66 |
| Table 21: | Time to Recovery by Treatment Group within Subgroups – As Treated Population | 66 |
| Table 22: | Time to Recovery by Treatment Group and Randomized Disease Severity: Readmittance Sensitivity Analysis – ITT Population | 66 |
| Table 23: | Time to Recovery by Treatment Group and Randomized Disease Severity: Medications of Interest Sensitivity Analysis – ITT Population | 66 |
| Table 24: | Summary of Recoveries and Deaths by Day 29 – ITT Population | 67 |
| Table 25: | Odds Ratio for Better (Lower) Clinical Status Score at Study Visit Day 15 by Treatment Using a Proportional Odds Model, Baricitinib + RDV Relative to Placebo + RDV – ITT Population | 68 |
| Table 26: | Odds Ratio for Better (Lower) Clinical Status Score at Study Visit Day 15 by Treatment Using a Proportional Odds Model, Baricitinib + RDV Relative to Placebo + RDV – As Treated Population | 69 |
| Table 27: | Time to Improvement on the 8-Point Ordinal Scale by Treatment Group | 70 |
| Table 28: | Time to Improvement on the 8-Point Ordinal Scale by Treatment Group: Modified Ordinal Scale | 70 |
| Table 29: | Time to Improvement by at least One Clinical Status Category on the 8-Point Ordinal Scale by Treatment Group within Subgroups – ITT Population | 70 |
| Table 30: | Time to Improvement by at least One Clinical Status Category on the 8-Point Ordinal Scale by Treatment Group within Subgroups – As Treated Population | 70 |
| Table 31: | Time to Improvement by at least Two Clinical Status Categories on the 8-Point Ordinal Scale by Treatment Group within Subgroups – ITT Population | 70 |
| Table 32: | Time to Improvement by at least Two Clinical Status Categories on the 8-Point Ordinal Scale by Treatment Group within Subgroups – As Treated Population | 70 |
| Table 33: | Clinical Status Scores by Treatment Group and Study Visit – ITT Population | 71 |
| Table 34: | Clinical Status Scores by Treatment Group and Study Visit – As Treated Population | 71 |
| Table 35: | Summary of Clinical Status Score by Treatment Group and Study Visit – ITT Population | 72 |
| Table 36: | Summary of Clinical Status Score by Treatment Group and Study Visit – As Treated Population | 72 |
| Table 37: | Time to Discharge or to a NEWS of < 2 by Treatment Group | 73 |

| Table 38: | Time to Discharge or to a NEWS of $\leq 2$ by Treatment Group within Subgroups – ITT Population. | 73 |
|---|---|---|
| Table 39: | Time to Discharge or to a NEWS of $\leq$ 2 by Treatment Group within Subgroups – As Treated Population | 73 |
| Table 40: | Summary of NEWS by Treatment Group and Study Visit – ITT Population | 74 |
| Table 41: | Summary of NEWS by Treatment Group and Study Visit – As Treated Population | 74 |
| Table 42: | Oxygen Use by Treatment Group | 75 |
| Table 43: | Oxygen Use by Treatment Group within Subgroups | 76 |
| Table 44: | Non-invasive Ventilation/High-Flow Oxygen Use by Treatment Group | 76 |
| Table 45: | Non-invasive Ventilation/High-Flow Oxygen Use by Treatment Group within Subgroups | 76 |
| Table 46: | Ventilation/ECMO Use by Treatment Group | 76 |
| Table 47: | Ventilation/ECMO Use by Treatment Group within Subgroups | 76 |
| Table 48: | Hospitalization by Treatment Group | 77 |
| Table 49: | Hospitalization by Treatment Group within Subgroups | 77 |
| Table 50: | Categorical Demographic and Baseline Characteristics by Randomized Disease Severity and Treatment Group – ITT Population | 78 |
| Table 51: | Continuous Demographic and Baseline Characteristics by Randomized Disease Severity and Treatment Group – ITT Population | 80 |
| Table 52: | Summary of Subjects with Pre-Existing Medical Conditions Treatment<br>Group - As Treated Population | 82 |
| Table 53: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification, Actual Disease Severity, and Treatment Group – As Treated Population | 83 |
| Table 54: | Number and Percentage of Subjects Reporting Use of Medications of Interest by Actual Disease Severity, and Treatment Group – As Treated Population | 84 |
| Table 55: | Use of Medications of Interest by Study Day, Actual Disease Severity, and Treatment Group – As Treated Population | 85 |
| Table 56: | Overall Summary of Adverse Events – As Treated Population | 86 |
| Table 57: | Subject-Level Rates of Adverse Events and Differences between Treatment<br>Groups – As Treated Population | 88 |
| Table 58: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - As Treated Population | 89 |

| Table 59: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Moderate Disease Severity, As Treated Population | 89 |
|---|---|---|
| Table 60: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Severe Disease Severity, As Treated Population | 89 |
| Table 61: | Treatment-Emergent Renal Adverse Events by Preferred Term and Treatment Group – As Treated Population | 90 |
| Table 62: | Treatment-Emergent Hepatic Adverse Events by Preferred Term and Treatment Group – As Treated Population | 90 |
| Table 63: | Related Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group - As Treated Population | 90 |
| Table 64: | Deaths by Day 15 or Day 29 by Treatment Group and Randomized Disease<br>Severity – ITT Population | 91 |
| Table 65: | Deaths by Day 15 or Day 29 by Treatment Group and Actual Disease<br>Severity – As Treated Population | 91 |
| Table 66: | Time to Death through Day 15 and 29 by Treatment Group and Randomized Disease Severity – ITT Population | 92 |
| Table 67: | Time to Death through Day 15 and 29 by Treatment Group and Actual Disease Severity – As Treated Population | |
| Table 68: | Time to Death through Day 15 and 29 by Treatment Group within Subgroups – ITT Population | 92 |
| Table 69: | Time to Death through Day 15 and 29 by Treatment Group: Medications of Interest Sensitivity Analysis – ITT Population | 92 |
| Table 70: | Time to Death through Day 15 and 29 by Treatment Group: Interaction Modeling – ITT Population | 92 |
| Table 71: | Time to Death through Day 15 and 29 by Treatment Group: Restricted Mean Survival Time Analysis – ITT Population | 94 |
| Table 72: | Subjects Experiencing Grade 3 or 4 AEs and SAEs through Day 29 by Treatment Group and Actual Disease Severity – As Treated Population | 95 |
| Table 73: | Analysis of Time to Death, SAEs, or Grade 3 or 4 AEs by Treatment Group – As Treated Population | |
| Table 74: | Infections by Treatment Group – As Treated Population, Moderate Disease Severity | |
| Table 75: | Opportunistic Infections by Treatment Group – As Treated Population, Moderate Disease Severity | |
| Table 76: | Infections by Treatment Group – As Treated Population, Severe Disease Severity | 97 |

| Table 77: | Opportunistic Infections by Treatment Group – As Treated Population, Severe Disease Severity |
|---|---|
| Table 78: | Infections by Treatment Group – As Treated Population, All Subjects97 |
| Table 79: | Opportunistic Infections by Treatment Group – As Treated Population, All Subjects |
| Table 80: | Abnormal Laboratory Results of Grade 3 or 4 by Parameter, Maximum Severity, Time Point, and Treatment Group – As Treated Population98 |
| Table 81: | Abnormal Laboratory Results of Grade 3 or 4 by Parameter, Maximum Severity, Time Point, and Treatment Group – Moderate Disease Severity, As Treated Population |
| Table 82: | Abnormal Laboratory Results of Grade 3 or 4 by Parameter, Maximum Severity, Time Point, and Treatment Group – Severe Disease Severity, As Treated Population |
| Table 83: | Treatment-Emergent Laboratory Abnormalities - As Treated Population99 |
| Table 84: | Summary Statistics of Laboratory Results by Parameter, Study Visit Day, and Treatment Group – As Treated Population |
| Table 85: | Summary Statistics of Laboratory Results by Parameter, Study Visit Day, and Treatment Group – Moderate Disease Severity, As Treated Population100 |
| Table 86: | Summary Statistics of Laboratory Results by Parameter, Study Visit Day, and Treatment Group – Severe Disease Severity, As Treated Population100 |

**Table 1:** Ineligibility Summary of Screen Failures

| | n <sup>a</sup> | % b |
|---|---|---|
| Total number of subjects failing any eligibility criterion or were eligible but not enrolled | X | 100 |
| Number of subjects failing any eligibility criterion | X | XX |
| Any inclusion criterion | X | XX |
| [inclusion criterion 1] | X | XX |
| [inclusion criterion 2] | X | XX |
| [inclusion criterion 3] | X | XX |
| Any exclusion criterion | X | XX |
| [exclusion criterion 1] | X | XX |
| [exclusion criterion 2] | X | XX |
| [exclusion criterion 3] | X | XX |
| | X | XX |
| b | Number of subjects failing any eligibility criterion Any inclusion criterion inclusion criterion 1] inclusion criterion 2] inclusion criterion 3] Any exclusion criterion exclusion criterion 1] exclusion criterion 2] | Number of subjects failing any eligibility criterion Any inclusion criterion X Inclusion criterion 2] X Inclusion criterion 3] Any exclusion criterion X Exclusion criterion 1] X Exclusion criterion 2] X Exclusion criterion 3] X Exclusion criterion 3] X Exclusion criterion 3] X Exclusion criterion 3] X Exclusion criterion 3] |

<sup>&</sup>lt;sup>b</sup> Denominator for percentages is the total number of screen failures.

# Programming Note:

Subjects who are eligible but not enrolled will be counted in the denominator.

Table 2: Analysis Population Eligibilities by Treatment Group and Randomized Disease Severity

| | | Baricitini | ib + RDV | Placebo - | + RDV | All Subjects | |
|---|---|---|---|---|---|---|---|
| Analysis | | Moderate | Severe | Moderate | Severe | Moderate | Severe |
| Population | Inclusion / Reason for Exclusion | n | n | n | n | n | n |
| Intention-to-Treat<br>Population | Included in Population <sup>1</sup> | X | Х | х | х | х | Х |
| As Treated | Included in Population <sup>2</sup> | х | Х | x | X | х | X |
| Population | Excluded from Population <sup>1</sup> | х | х | x | X | х | X |
| | Did Not Receive Dose of<br>Baricitinib/Placebo <sup>1</sup> | X | Х | Х | X | Х | X |

Counts are the numbers of subjects randomized to the specified treatment group and randomized disease severity stratum.

## **Programming Notes:**

If at least one subject received the incorrect treatment, then a footnote will be added which reads "XX subject[s] [was/were] randomized to [insert randomized treatment] but was administered [insert actual treatment]. In addition, a row under "Included in Population" and "Excluded from Population" will be added for the As Treated Population section with the label "Randomized to [insert randomized treatment] but administered [insert actual treatment]."

If at least one subject was randomized to the incorrect disease severity stratum then a separate table will be generated which classifies subjects by their actual disease severity. The title of the table will be: "Analysis Population Eligibilities by Treatment Group and Actual Disease Severity". If needed, the table format used for ACTT-1 will be used.

<sup>&</sup>lt;sup>2</sup> Counts are the numbers of subjects in the randomized disease severity stratum who received the specified treatment.

Table 3: Subject Disposition by Treatment Group and Randomized Disease Severity – ITT Population

| | В | | ib + RD'<br>=X) | V | ] | | + RDV<br>=X) | All Subjects (N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Moderate<br>(N=X) | | Sev<br>(N= | - | Moderate<br>(N=X) | | Severe<br>(N=X) | | Moderate<br>(N=X) | | | ere<br>=X) |
| Subject Disposition | n/N | % | n/N | % | n/N | % | n/N | % | n/N | % | n/N | % |
| Randomized | x/x | 100 | x/x | 100 | x/x | 100 | x/x | 100 | x/x | 100 | x/x | 100 |
| Completed Follow-up (Study Day 1) –<br>Hospitalized Subjects in Study | x/x | xx | x/x | XX | x/x | xx | x/x | XX | x/x | XX | x/x | XX |
| Ordinal Scale Data Available | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| NEWS Data Scale Data Available | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Safety Laboratory Blood Draw | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| OP Swab Collection | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| PCR Assays Blood Draw | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Secondary Research Blood Draw | x/x | XX | x/x | xx | x/x | XX | x/x | XX | x/x | xx | x/x | xx |
| Continue for Days 3, 5, 8, 11 for hospitalized subje | cts. | | | | | | | | | | | |
| Completed Follow-up (Study Day 15) – All Subjects in Study | x/x | xx | x/x | XX | x/x | xx | x/x | XX | x/x | XX | x/x | XX |
| Ordinal Scale Data Available | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| NEWS Data Scale Data Available | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Safety Laboratory Blood Draw | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| OP Swab Collection | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Secondary Research Blood Draw | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Completed Follow-up (Study Day 22) – All Subjects in Study | x/x | xx | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Ordinal Scale Data Available | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| NEWS Data Scale Data Available (Inpatient Subjects Only) | x/x | xx | x/x | XX | x/x | xx | x/x | XX | x/x | XX | x/x | XX |
| Completed Follow-up (Study Day 29) – All Subjects in Study | x/x | xx | x/x | Xx | x/x | xx | x/x | XX | x/x | XX | x/x | XX |
| Ordinal Scale Data Available | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| NEWS Data Scale Data Available | x/x | xx | x/x | xx | x/x | xx | x/x | XX | x/x | XX | x/x | xx |
| Safety Laboratory Blood Draw | x/x | xx | x/x | XX | x/x | xx | x/x | XX | x/x | XX | x/x | xx |
| OP Swab Collection | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |
| Secondary Research Blood Draw | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX | x/x | XX |

N = Number of subjects enrolled and in study for visits 1, 15, 22 and 29 and the number of subjects hospitalized and in study for visits 3, 5, 8 and 11. Subjects that died or terminated from the study on or prior to the study visit are not included in the denominators.

**Table 4:** Treatment Compliance by Treatment Group

| | Baricitinib + RDV<br>(N=X) | | | P | lacebo + F<br>(N=X) | RDV | | l Subjec<br>(N=X) | ets | Proportion<br>Difference | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Disposition | n | % | 95%CIa | n | % | 95%CI | n | % | 95%CI | % | 95%CI |
| Received Remdesivir Prior to Enrollment | X | X | x.x, x.x | X | X | x.x, x.x | х | х | x.x, x.x | X | x.x, x.x |
| Received First On-Study Dose of Remdesivir | X | x | x.x, x.x | x | X | x.x, x.x | х | х | x.x, x.x | X | x.x, x.x |
| Received at least one Oral<br>Dose of Baricitinib/Placebo | X | x | x.x, x.x | x | х | x.x, x.x | x | x | x.x, x.x | X | x.x, x.x |
| Received all 10 Infusions of<br>Remdesivir | X | x | x.x, x.x | x | х | x.x, x.x | x | x | x.x, x.x | X | x.x, x.x |
| Received all 14 Oral Doses of<br>Barcitinib/Placebo | X | х | x.x, x.x | X | х | x.x, x.x | х | x | x.x, x.x | X | x.x, x.x |
| Received less than 10 Infusions of Remdesivir due to Discharge | X | х | x.x, x.x | X | x | x.x, x.x | x | х | x.x, x.x | X | x.x, x.x |
| Received less than 10 Infusions of Remdesivir due to Death | X | X | x.x, x.x | X | х | x.x, x.x | x | х | x.x, x.x | X | x.x, x.x |
| Received less than 14 doses of<br>Baricitinib/Placebo due to<br>Discharge | X | Х | x.x, x.x | X | x | x.x, x.x | х | x | x.x, x.x | x | x.x, x.x |
| Received less than 14 doses of<br>Baricitinib/Placebo due to<br>Death | X | x | x.x, x.x | X | x | x.x, x.x | x | х | x.x, x.x | X | x.x, x.x |
| Had Any Infusions of<br>Remdesivir Halted or Slowed | X | x | x.x, x.x | X | х | x.x, x.x | х | х | x.x, x.x | X | x.x, x.x |
| Had Any Oral Doses of<br>Baricitinib/Placebo Modified | X | X | x.x, x.x | x | x | x.x, x.x | x | х | x.x, x.x | x | x.x, x.x |
| Missed Any Maintenance Dose of Remdesivir | X | X | x.x, x.x | X | X | x.x, x.x | X | х | x.x, x.x | x | x.x, x.x |
| Missed Any Oral Dose of<br>Baricitinib/Placebo | X | X | x.x, x.x | x | х | x.x, x.x | х | х | x.x, x.x | x | x.x, x.x |

N = Number of subject enrolled

#### **Programming Notes:**

Received On-Study Dose: Subjects received the first treatment: EC.ECTPT = DOSE 1.

Infusions/doses are counted as "Received" even if they are halted/slowed/modified.

Had any infusions halted or slowed: EC.ECADJ is not missing through day 10 or through discharge from hospital or death.

Missed any maintenance dose: EC.ECOCCUR=N through day 10 or through discharge from hospital or death.

95% CI for proportions obtained by Clopper-Pearson:

<sup>95%</sup> CI for proportions obtained by Clopper-Pearson

<sup>95%</sup> CI for difference in proportions obtained by the exact method

```
proc freq;
        Table treatment*analysisvariable / binomial;
        ods output binomialcls=outputdsn;
run;

95% CI for difference in proportions obtained by the exact method:
proc freq;
        Table treatment*analysisvariable / riskdiff (cl=exact);
run;
```

Table 5: Subjects Reporting Prior Remdesivir Treatment by Randomized Disease Severity and Treatment Group – ITT Population

| | | ib + RDV<br>=X) | | o + RDV<br>=X) | All Subjects (N=X) | |
|---|---|---|---|---|---|---|
| Prior RDV Treatment Summary | Moderate<br>(N=X) | Severe<br>(N=X) | Moderate<br>(N=X) | Severe<br>(N=X) | Moderate<br>(N=X) | Severe<br>(N=X) |
| Received RDV Treatment Prior to Enrollment – n (%) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Number of Doses of RDV Received Prior to Enrollment | | | | | | |
| Number of Subjects with Data | X | х | X | х | х | х |
| Mean (STD) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| Median | X.X | X.X | X.X | X.X | X.X | X.X |
| IQR | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | X.X, X.X |
| Range (Min, Max) | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | X.X, X.X |
| N = Number of subjects in the ITT Population. | | l . | l . | l . | l. | I |

Table with similar format:

Table 6: Subjects Reporting Prior Remdesivir Treatment by Actual Disease Severity and Treatment Group – As Treated Population

Table 7: Distribution of Subject Specific Protocol Deviations by Category, Type, Treatment Group, and Randomized Disease Severity

| | | Baricitinib + RDV<br>(N=X) | | | | | | 00 + RDV<br>N=X) | All Subjects<br>(N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Moderate<br>(N=X) | | Severe<br>(N=X) | | Moderate<br>(N=X) | | Severe<br>(N=X) | | Moderate<br>(N=X) | | Sev<br>(N= | |
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Eligibility/enrollment | Any type | х | х | X | х | х | Х | х | х | X | X | х | X |
| | Did not meet inclusion criterion | х | X | Х | х | X | Х | х | Х | Х | X | Х | X |
| | Met exclusion criterion | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | ICF not signed prior to study procedures | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | Other | х | х | Х | х | х | х | х | х | Х | х | х | X |
| Treatment administration schedule | Any type | х | Х | Х | х | Х | х | х | Х | х | x | Х | X |
| | Out of window visit | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | Missed visit/visit not conducted | х | х | Х | х | х | х | х | х | Х | х | х | X |
| | Missed treatment administration | х | Х | х | х | Х | х | х | х | х | x | Х | X |
| | Delayed treatment administration | х | Х | Х | х | Х | х | х | Х | х | x | Х | X |
| | Other | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| Follow-up visit schedule | Any type | х | Х | Х | х | Х | х | х | Х | х | x | Х | X |
| | Out of window visit | х | х | Х | х | х | х | х | х | Х | х | х | X |
| | Missed visit/visit not conducted | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | Other | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| Protocol procedure/assessment | Any type | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | Incorrect version of ICF signed | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | Blood not collected | х | х | Х | х | х | х | х | х | Х | х | х | X |
| | Oropharyngeal swab not collected | х | Х | Х | х | Х | х | х | Х | Х | х | Х | X |
| | Other specimen not collected | х | Х | х | х | х | х | х | х | Х | x | х | X |
| | Specimen result not obtained | х | Х | х | х | х | х | х | х | Х | x | х | X |
| | Required procedure not conducted | х | Х | Х | х | Х | х | х | Х | X | X | Х | X |

| | | | | | Baricitinib + RDV<br>(N=X) | | | | | All Subjects<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Moderate<br>(N=X) | | Severe<br>(N=X) | | Moderate<br>(N=X) | | Severe<br>(N=X) | | Moderate<br>(N=X) | | | ere<br>=X) |
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| | Required procedure done incorrectly | x | x | Х | х | Х | Х | X | Х | Х | х | Х | X |
| | Study product temperature excursion | x | X | х | x | Х | х | X | Х | х | х | х | X |
| | Specimen temperature excursion | x | X | х | x | Х | х | X | Х | х | х | х | X |
| | Stratification error | x | X | х | x | Х | х | X | Х | х | х | х | X |
| | Other | x | X | Х | Х | Х | Х | x | Х | Х | х | Х | X |
| Treatment administration | Any type | x | X | Х | X | Х | Х | X | Х | Х | х | Х | X |
| | Required procedure done incorrectly | x | X | х | x | Х | х | X | Х | х | х | х | X |
| | Study product temperature excursion | x | X | Х | Х | Х | Х | x | Х | Х | х | Х | X |
| | Other | x | X | Х | Х | Х | Х | x | Х | Х | х | Х | X |
| Blinding policy/procedure | Any type | x | X | Х | Х | Х | Х | x | Х | Х | х | Х | X |
| | Treatment unblinded | X | X | х | х | х | х | x | х | х | х | х | X |
| | Other | X | Х | Х | Х | Х | х | х | Х | Х | Х | Х | X |
| N = number of subjects enrolled | | | 1 | | | | 1 | | | | | | |

Tables with similar format:

- Table 8: Distribution of Subject Specific Protocol Deviations by Category, Type, and Geographic Region
- Table 9: Distribution of Major Subject Specific Protocol Deviations by Category, Type, Treatment Group, and Randomized Disease

Severity

- Table 10: Distribution of Major Subject Specific Protocol Deviations by Category, Type, and Geographic Region
- Table 11: Distribution of Non-Subject Specific Protocol Deviations by Category and Type
- Table 12: Distribution of Non-Subject Specific Protocol Deviations by Category, Type, and Geographic Region
- Table 13: Distribution of Major Non-Subject Specific Protocol Deviations by Category and Type
- Table 14: Distribution of Major Non-Subject Specific Protocol Deviations by Category, Type, and Geographic Region

Programming Notes for Tables 8, Table 10, Table 12, and Table 14:

Geographic Region will be North America vs. Europe vs. Asia.

Table 15: Time to Recovery by Treatment Group and Randomized Disease Severity

| Analysis | | | | Median Time to Recovery | | Н | | |
|---|---|---|---|---|---|---|---|---|
| Population | Treatment Group | Disease Severity | n | Estimate | 95% CI | Estimate | 95% CI | P-value |
| ITT Population | Baricitinib + RDV (N=X) | Moderate | X | X.X | x.x, x.x | V VV | x.xx,<br>x.xx | |
| | Placebo + RDV (N=X) | | X | X.X | x.x, x.x | X.XX | | |
| | Baricitinib + RDV (N=X) | Severe | X | X.X | X.X, X.X | | x.xx, | |
| | Plaecbo + RDV (N=X) | | X | X.X | X.X, X.X | X.XX | x.xx | |
| | Baricitinib + RDV (N=X) | Any Severity | X | X.X | x.x, x.x | | x.xx, | 0 |
| | Placebo + RDV (N=X) | | X | X.X | x.x, x.x | X.XX | x.xx | 0.xxx |

Repeat for the As Treated Population.

Tables with similar format:

Table 16: Time to Recovery by Treatment Group and Randomized Disease Severity: Fine-Gray, Covariate-Adjusted, and Interaction Modeling

Table 17: Time to Recovery by Treatment Group and Baseline Ordinal Score: Fine-Gray and Interaction Modeling

Programming Notes for Table 16 and Table 17:

For both tables, the median time columns will be excluded.

The "Analysis Population" column will be replaced by a "Model" column. For the Fine-Gray estimates, the column will display "Fine-Gray", for the covariate-adjusted model, the column will display "Covariate-Adjusted", and for the interaction models (Table 16), the columns will display, respectively, for the three models to be run:

- "Treatment-Severity Interaction (Randomized Severity)"
- "Treatment-Severity Interaction (Actual Severity)"

For the interaction models, the p-value for the interaction term will be provided in a footnote reading "The p-value for the treatment by [randomized/actual] disease severity interaction term was 0.xxxx.".

For the covariate-adjusted model, a cox model will be run with age, duration of symptoms prior to enrollment, baseline d-dimer, and baseline CRP values included as continuous covariates.

For Table 17, the interaction model column will display "Baseline Ordinal Score Interaction". For the interaction models, the p-value for the interaction term will be provided in a footnote reading "The p-value for the treatment by baseline ordinal score interaction term was 0.xxxx.".

N= Number of subjects in the specified treatment group, disease severity, and analysis population.

n = Number of recovered subjects.

HR is the ratio of the hazard of recovery in each treatment group estimated from the Cox model. The ratio is Baricitinib + RDV to Placebo + RDV.

HR for the 'Any Severity' group is the hazard ratio from the stratified Cox Model.

P-value calculated using the stratified log-rank test

Table 18: Time to Recovery by Treatment Group and Disease Severity: Restricted Mean Survival Time Analysis – ITT Population

| Analysis | | Randomized | | Restricted Me<br>Tin | | Difference | |
|---|---|---|---|---|---|---|---|
| Population Population | Treatment Group | Disease Severity | n | Estimate | 95% CI | Estimate | 95% CI |
| ITT Population | Baricitinib + RDV (N=X) | Moderate | X | X.X | x.x, x.x | | x.xx,<br>x.xx |
| | Placebo + RDV (N=X) | | X | X.X | x.x, x.x | X.XX | |
| | Baricitinib + RDV (N=X) | Severe | X | X.X | x.x, x.x | V VV | xx x.xx,<br>x.xx |
| | Plaecbo + RDV (N=X) | | X | X.X | x.x, x.x | X.XX | |
| | Baricitinib + RDV (N=X) | Any Severity | X | X.X | x.x, x.x | V VV | x.xx, |
| | Plaecbo + RDV (N=X) | | X | X.X | x.x, x.x | X.XX | x.xx |

Repeat for the As Treated Population.

#### **Programming Notes:**

Within a severity stratum:

```
proc lifetest data=enrevent plots=(rmst) method=breslow rmst(cl);
by stratum;
time evntday * Censor(1);
strata trtcode /diff=all;
ods output rmst=rmst;
run;
```

Stratified by disease severity ("Any Severity" row).

```
proc lifetest data=enrevent plots=(rmst) method=breslow rmst(cl);
time evntday * Censor(1);
strata trtcode CRSEVERE /diff=all;
ods output rmst=rmst;
run;
```

**Table 19:** Time to Recovery by Treatment Group within Prior RDV Treatment Subgroups

| | | Prior RDV | | Median Time | to Recovery | HR | |
|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Treatment Group | Treatment<br>Subgroup | n | Estimate | 95% CI | Estimate | 95% CI |
| ITT Population | Baricitinib + RDV (N=X) | No Prior | х | X.X | x.x, x.x | | x.xx,<br>x.xx |
| | Placebo + RDV (N=X) | Treatment | х | X.X | x.x, x.x | X.XX | |
| | Baricitinib + RDV (N=X) | Any Prior<br>Treatment | х | X.X | x.x, x.x | | x.xx,<br>x.xx |
| | Plaecbo + RDV (N=X) | | Х | x.x | x.x, x.x | X.XX | |

Repeat for the As Treated Population.

N= Number of subjects in the specified treatment group, disease severity, and analysis population.

n = Number of recovered subjects.

Difference is the difference in the restricted mean recovery time between Baricitinib + RDV and Placebo + RDV.

N= Number of subjects in the specified treatment group, disease severity, and analysis population.

n = Number of recovered subjects.

HR is the ratio of the hazard of recovery in each treatment group estimated from the Cox model. The ratio is Baricitinib + RDV to Placebo + RDV.

Additional tables with similar format as Table 15:

- **Table 20:** Time to Recovery by Treatment Group within Subgroups ITT Population
- Table 21: Time to Recovery by Treatment Group within Subgroups As Treated Population
- Table 22: Time to Recovery by Treatment Group and Randomized Disease Severity: Readmittance Sensitivity Analysis ITT Population
- Table 23: Time to Recovery by Treatment Group and Randomized Disease Severity: Medications of Interest Sensitivity Analysis ITT Population

Programming Notes for Tables 20 and 21:

The "Disease Severity" and "Analysis Population" columns will be removed. A "Subgroup" column will be inserted to the left of the "Treatment Group" column. These tables will not display the "Any..." rows. For the analysis controlling for age, symptom duration, d-dimer, and CRP values as continuous covariates, the elements for the "Subgroup" column will state "Baseline Predictors as Continuous Covariates". The elements for the "n" and "Median Time to Recovery" columns will display "-". P-values will not be included in these tables.

Programming Notes for Tables 22 and 23:

P-values will not be included in these tables.

Table 22 will include a column to the left of the "n" column titled "m". The corresponding footnote will read "m = Number of subjects readmitted for COVID-19." Table 11 will include the following footnote: "In this analysis, subjects that recover and are subsequently readmitted for COVID-19 are censored at 28 days".

Table 23 will include a column to the left of the "n" column titled "m". The corresponding footnote will read "m = Number of subjects reporting use of the medication of interest." For Table 12, the "Analysis Population" column will be replaced by a column labeled "Medication of Interest". Separate models will be fit for the following categories of medications (see Section 6.4):

- Any Medication of Interest
- Hydroxychloroquine/Chloroquine
- Corticosteroids
- Anti-Inflammatory Drugs

The table will include the following footnote: "In this analysis, subjects that reported use of the specified medications of interest (Section 6.4 of the SAP) are censored at time of medication receipt."

**Table 24:** Summary of Recoveries and Deaths by Day 29 – ITT Population

| Grouping | | | Reco | vered | Did Not | Recover | Dea | nths | Not Reco | |
|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Subgroup | Treatment Group | n | % | n | % | n | % | n | % |
| Disease<br>Severity | Moderate | Baricitinib + RDV (N=X) | X | X | x | X | X | X | X | X |
| | | Placebo + RDV (N=X) | X | X | x | X | X | X | X | X |
| | Severe | Baricitinib + RDV (N=X) | X | X | X | X | X | X | X | X |
| | | Placebo + RDV (N=X) | X | X | X | X | X | Х | Х | X |
| | Any Severity | Baricitinib + RDV (N=X) | X | X | х | X | X | Х | X | X |
| | | Placebo + RDV (N=X) | X | X | Х | Х | X | х | X | X |

Repeat for duration of symptoms categories in Section 6.4

N= Number of subjects in the ITT Population.

Programming Note: For the categories of "Recovered", "Did Not Recover" and "Deaths", subjects who recover but subsequently die will be classified under "Recovered" and "Deaths". If there are cases of this, a footnote will be added that states "Counts of recoveries and deaths include X subjects who recovered but subsequently died."

Table 25: Odds Ratio for Better (Lower) Clinical Status Score at Study Visit Day 15 by Treatment Using a Proportional Odds Model, Baricitinib + RDV Relative to Placebo + RDV – ITT Population

| | | Odds | Odds Ratio | |
|---|---|---|---|---|
| Analysis/Subgroup | Treatment Group | Estimate | 95% CI | P-value |
| | Main Analysis of Key Seco | ndary Endpoint | | |
| Analysis of Key Secondary Endpoint <sup>1</sup> | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | 0.xxx |
| | Subgroup Analyses of Key Se | econdary Endpoint | | |
| [Repeat for each Section 6.4 | Baricitinib + RDV (N=X) | | | |
| subgroups] | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| | Medications of Interest Sen | sitivity Analyses | | |
| Any Medication of Interest | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| Hydroxychloroquine/Chloroquine | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| Corticosteroids | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| Anti-Inflammatory Drugs | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| | Covariate-Adjuste | d Model | | |
| Covariate-Adjusted | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| | Interaction Mo | dels | | |
| Treatment-Severity Interaction | Baricitinib + RDV (N=X) | | | |
| | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| Treatment-Baseline Ordinal Score | Baricitinib + RDV (N=X) | | | |
| Interaction | Placebo + RDV (N=X) | x.xx | x.xx, x.xx | |
| <sup>1</sup> Analysis of key secondary endpoir | nt using the full As Treated Populat | ion with disease severit | y as a model covaria | ite. |

Programming Note: P-value of treatment comparison will only be displayed for the main analysis. For the interaction models, the p-value for the interaction term will be provided in a footnote reading "The p-value for the treatment by disease severity interaction term was 0.xxxx.".

For the covariate-adjusted model, the model will be run with age, duration of symptoms prior to enrollment, baseline d-dimer, and baseline CRP values included as continuous covariates.

Table with similar format:

Table 26: Odds Ratio for Better (Lower) Clinical Status Score at Study Visit Day 15 by Treatment Using a Proportional Odds Model, Baricitinib + RDV Relative to Placebo + RDV – As Treated Population

Programming Note: P-value of treatment comparison will only be displayed for the main analysis. For the interaction models, the p-value for the interaction term will be provided in a footnote reading "The p-value for the treatment by disease severity interaction term was 0.xxxx."

**Table 27:** Time to Improvement on the 8-Point Ordinal Scale by Treatment Group

| Analysis | | Median Time | | Н | | | |
|---|---|---|---|---|---|---|---|
| Population <b>Population</b> | Treatment Group | n | Estimate | 95% CI | Estimate | 95% CI | P-value |
| Improvement by at least One Category | | | | | | | |
| ITT Population | Baricitinib + RDV (N=X) | x | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | х | X.X | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |
| As Treated | Baricitinib + RDV (N=X) | х | X.X | x.x, x.x | | | |
| Population | Placebo + RDV (N=X) | х | X.X | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |
| | Imp | rovement b | y at least Two C | Categories | | | |
| ITT Population | Baricitinib + RDV (N=X) | x | X.X | x.x, x.x | | | |
| | Placebo + RDV (N=X) | х | X.X | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |
| As Treated | Baricitinib + RDV (N=X) | x | X.X | x.x, x.x | | | |
| Population | Placebo + RDV (N=X) | x | X.X | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |

N = Number of subjects in the specified treatment group and analysis population.

#### Tables with similar format:

- Table 28: Time to Improvement on the 8-Point Ordinal Scale by Treatment Group: Modified Ordinal Scale
- Table 29: Time to Improvement by at least One Clinical Status Category on the 8-Point Ordinal Scale by Treatment Group within Subgroups ITT Population
- Table 30: Time to Improvement by at least One Clinical Status Category on the 8-Point Ordinal Scale by Treatment Group within Subgroups As Treated Population
- Table 31: Time to Improvement by at least Two Clinical Status Categories on the 8-Point Ordinal Scale by Treatment Group within Subgroups ITT Population
- Table 32: Time to Improvement by at least Two Clinical Status Categories on the 8-Point Ordinal Scale by Treatment Group within Subgroups As Treated Population

#### Programming notes for Table 28:

The table will include the footnote: This analysis used the modified version of the ordinal scale where the categories "Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care" and "Not hospitalized, no limitations on activities" were classified together and given a score of 2 while the category "Not hospitalized, limitation on activities" was given the score 3."

Programming notes for Tables 29, Table 30, Table 31, Table 32: Instead of the "Analysis Population" column, columns titled "Subgroup Category" and "Subgroup" will be to the left of Treatment Group. Rows will be generated for each subgroup. Since the One and Two Category improvement outcomes are presented separately in these tables, the spanned row of "Improvement by at least XXX" will not be displayed in these tables.

n = Number of subjects with improvement.

HR is the ratio of the hazard of improvement in each treatment group estimated from the Cox model. The ratio is Baricitinib + RDV to Placebo + RDV.

P-value calculated using the Log-rank test

Table 33: Clinical Status Scores by Treatment Group and Study Visit – ITT Population

| | Ordinal Scale Measure | | Baricitinib + RDV<br>(N=X) | | | Placebo + RDV<br>(N=X) | | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit | | | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Day 1 | Death at or before Study Visit (8) | Х | х | x.x, x.x | x | х | x.x, x.x | X | х | x.x, x.x |
| | Hospitalized, on invasive mechanical ventilation or ECMO (7) | х | х | x.x, x.x | х | х | x.x, x.x | x | х | x.x, x.x |
| | Hospitalized, on non-invasive ventilation or high flow oxygen devices (6) | Х | х | x.x, x.x | х | х | x.x, x.x | х | х | x.x, x.x |
| | Hospitalized, requiring supplemental oxygen (5) | Х | х | x.x, x.x | х | x | x.x, x.x | X | х | x.x, x.x |
| | Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise) (4) | х | х | x.x, x.x | х | х | x.x, x.x | X | x | x.x, x.x |
| | Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (3) | х | х | x.x, x.x | х | X | x.x, x.x | x | х | x.x, x.x |
| | Not hospitalized, limitation on activities and/or requiring home oxygen (2) | Х | х | x.x, x.x | x | х | x.x, x.x | x | х | x.x, x.x |
| | Not hospitalized, no limitations on activities (1) | Х | х | x.x, x.x | x | х | x.x, x.x | x | х | x.x, x.x |
| | No clinical status score reported – Hospitalized subjects | х | х | x.x, x.x | x | х | x.x, x.x | x | х | x.x, x.x |
| | No clinical status score reported – Discharged subjects | X | x | x.x, x.x | X | X | x.x, x.x | X | х | x.x, x.x |

[Repeat for Study Visit Days 3, 5, 8, 11, 15, 22, and 29]

# Programming Notes:

If necessary, a row for "No clinical status score reported – Completed study without reporting score" will be added as the last row for each day.

#### Table with similar format:

## Table 34: Clinical Status Scores by Treatment Group and Study Visit – As Treated Population

N = Number of Subject in the ITT Population.

n = Number of subjects who reported the respective score

<sup>95%</sup> CI calculated using Wilson Cis

Table 35: Summary of Clinical Status Score by Treatment Group and Study Visit – ITT Population

| Study Visit | Statistic | Baricitinib + RDV<br>(N=X) | Placebo + RDV<br>(N=X) | All Subjects<br>(N=C) |
|---|---|---|---|---|
| Baseline | Number of reported clinical scores | X | X | X |
| | Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Median | X.X | X.X | X.X |
| | Range (Min, Max) | x, x | x, x | x, x |
| Day 3 | Number of reported clinical scores | Х | X | X |
| | Mean (SD) | x.x(x.x) | x.x (x.x) | x.x (x.x) |
| | Median | X.X | X.X | X.X |
| | Range (Min, Max) | x, x | x, x | x, x |
| | Change from Baseline Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) |

Continue for Days 5, 8, 11, 15, 22, 29

Table with similar format:

Table 36: Summary of Clinical Status Score by Treatment Group and Study Visit – As Treated Population

N = Number of subjects in the ITT Population.

SD = Standard deviation.

Missing values were imputed using Last Observation Carried Forward. Clinical scores of 8 were carried forward from the date of death for subjects who died.
Table 37: Time to Discharge or to a NEWS of  $\leq 2$  by Treatment Group

| Analysis | | | Media | ın Time | НЕ | ₹ | |
|---|---|---|---|---|---|---|---|
| Population | Treatment Group | nª | Estimate | 95% CI | Estimate | 95% CI | P-value |
| ITT Population | Baricitinib + RDV (N=X) | X | X.X | x.x, x.x | | | |
| | Placebo + RDV (N=X) | X | X.X | x.x, x.x | X.XX | x.xx, x.xx | X.XXX |
| As Treated | Baricitinib + RDV (N=X) | X | X.X | x.x, x.x | | | |
| Population | Placebo + RDV (N=X) | Х | X.X | x.x, x.x | X.XX | x.xx, x.xx | X.XXX |

N= Number of subjects in the specified treatment group and analysis population.

Table 38: Time to Discharge or to a NEWS of  $\leq 2$  by Treatment Group within Subgroups – ITT

**Population** 

Table 39: Time to Discharge or to a NEWS of  $\leq 2$  by Treatment Group within Subgroups – As

**Treated Population** 

Programming notes for Tables 38-39: "Subgroup Category" and "Subgroup" columns will replace the "Analysis Population" column to the left of "Treatment Group". Rows will be repeated for each subgroup. P-values will not be displayed in these tables.

n = Number of subjects who discharged or had a NEWS of  $\leq$  2 prior to Day 29.

HR is the ratio of the hazard of discharge or NEWS of  $\leq 2$  in each treatment group estimated from the Cox model. The ratio is Baricitinib + RDV to Placebo + RDV. P-value calculated using the Log-rank test

Table 40: Summary of NEWS by Treatment Group and Study Visit – ITT Population

| Study<br>Visit | Statistic | Baricitinib + RDV<br>(N=X) | Placebo + RDV<br>(N=X) | All Subjects<br>(N = X) |
|---|---|---|---|---|
| Baseline | n | Х | X | X |
| | Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Median | X.X | X.X | X.X |
| | Range (Min, Max) | X, X | X, X | x, x |
| Day 3 | n | Х | Х | X |
| | Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Median | X.X | X.X | X.X |
| | Range (Min, Max) | X, X | X, X | x, x |
| | n <sup>a</sup> | Х | Х | X |
| | Change from Baseline Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) |

[Repeat for Study Visit Days 5, 8, 11, 15, 22, 29 and Change from Baseline at each]

### Table with similar format:

Table 41: Summary of NEWS by Treatment Group and Study Visit – As Treated Population

n = Number of subjects with an assessment at both baseline and the time point being summarized.

n<sup>a</sup> = Number of subjects with an assessment at both baseline and the time point being summarized.

SD = Standard deviation.

**Table 42:** Oxygen Use by Treatment Group

| | | | Treatment | Group |
|---|---|---|---|---|
| <b>Analysis Population</b> | Oxygen Use | Statistic | Baricitinib + RDV | Placebo + RDV |
| ΓΤ Population | | On Oxygen at Bas | eline (N = x) | |
| | Days on Oxygen (Including | N | X | х |
| | imputations for subjects who died) | Q1 | X.X | x.x |
| | | Median | X.X | X.X |
| | | Q3 | X.X | X.X |
| | Days of Oxygen (Among subjects | N | X | x |
| | who did not die) | Q1 | X.X | x.x |
| | | Median | X.X | x.x |
| | | Q3 | X.X | x.x |
| | | Not on Oxygen at Ba | aseline $(N = x)$ | |
| | New Oxygen Use | N | X | x |
| | | n | X | x |
| | | Incidence Rate | X.X | x.x |
| | | Incidence Rate CI | X.X, X.X | x.x, x.x |
| | Days on Oxygen (Including | N | X | x |
| | imputations for subjects who died) | Q1 | X.X | x.x |
| | | Median | X.X | x.x |
| | | Q3 | X.X | x.x |
| | Days of Oxygen (Among subjects | N | X | X |
| | who did not die) | Q1 | X.X | X.X |
| | | Median | X.X | X.X |
| | | Q3 | X.X | X.X |

N = Number of subjects in the specified analysis population and oxygen use category.

# Programming Notes:

For the "Days on Oxygen" statistics within the "Not on Oxygen at Baseline" subgroup, only summarize days for subjects who reported new use.

Q1 and Q3 are the first and third quartiles, respectively.

- **Table 43:** Oxygen Use by Treatment Group within Subgroups
- Table 44: Non-invasive Ventilation/High-Flow Oxygen Use by Treatment Group
- Table 45: Non-invasive Ventilation/High-Flow Oxygen Use by Treatment Group within Subgroups
- **Table 46:** Ventilation/ECMO Use by Treatment Group
- **Table 47:** Ventilation/ECMO Use by Treatment Group within Subgroups

Programming notes for Table 43, Table 45, Table 47: "Analysis Population" will be replaced by "Grouping Variable" column. Summaries will only be generated for ITT population.

**Table 48:** Hospitalization by Treatment Group

| | | | Treatment | Group |
|---|---|---|---|---|
| <b>Analysis Population</b> | Summary | Statistic | Baricitinib + RDV | Placebo + RDV |
| ITT Population | Number of Subjects | N | X | X |
| | Days of Hospitalization | Q1 | X.X | X.X |
| | | Median | X.X | X.X |
| | | Q3 | X.X | X.X |
| | Incidence of Readmittance | N | X | X |
| | | Percentage | X | X |
| | | Percentage CI | x.x, x.x | x.x, x.x |

Continue for As Treated Population....

Table with similar format:

# **Table 49:** Hospitalization by Treatment Group within Subgroups

Programming notes for Table 49: "Analysis Population" will be replaced by "Grouping Variable" column. Summaries will only be generated for ITT population

N = Number of subjects in the specified analysis population.

Q1 and Q3 are the first and third quartiles, respectively.

Denominator of readmittance percentages is the number of subjects in the specific analysis population.

Table 50: Categorical Demographic and Baseline Characteristics by Randomized Disease Severity and Treatment Group – ITT Population

| | | | В | aricitini | ib + RD | V | | | | Placebo | + RDV | , | | | | All Su | bjects | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | lerate<br>=X) | | vere<br>=X) | | bjects<br>=X) | | erate<br>=X) | | vere<br>=X) | | bjects<br>=X) | | lerate<br>=X) | | vere<br>=X) | | ıbjects<br>=X) |
| <b>Demographic Category</b> | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | X | X | X | X | X | X | X | х | X | X | X | X | x | X | X | X | X | X |
| | Female | X | X | X | X | X | X | X | x | X | X | x | X | x | X | X | X | x | X |
| Ethnicity | Not Hispanic or Latino | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | x | X |
| | Hispanic or Latino | X | X | X | X | X | X | X | x | X | X | x | X | x | X | X | X | x | X |
| | Not Reported | X | X | X | X | X | X | X | X | X | X | X | X | х | Х | Х | X | x | X |
| | Unknown | х | х | x | x | х | х | х | х | х | х | х | X | х | х | х | х | х | х |
| Race | American Indian or Alaska<br>Native | X | x | X | X | х | х | x | х | X | X | x | х | х | х | х | х | x | X |
| | Asian | X | X | X | X | X | X | X | x | X | X | x | X | X | X | X | X | x | X |
| | Native Hawaiian or Other<br>Pacific Islander | X | х | х | х | х | Х | х | х | Х | Х | х | х | х | Х | х | х | х | х |
| | Black or African American | X | X | X | X | X | X | X | x | X | X | x | X | x | X | X | X | x | X |
| | White | x | x | x | x | X | x | х | х | x | X | x | X | х | x | x | x | x | x |
| | Multi-Racial | X | х | х | х | х | X | х | х | х | X | х | X | х | Х | х | х | х | х |
| | Unknown | х | х | x | X | X | х | х | х | х | X | х | X | х | х | x | х | х | х |
| Geographic Region | Region 1 | х | х | x | X | X | х | х | х | х | X | х | X | х | х | x | х | х | х |
| | Continue for all region categorizations | х | х | х | х | х | Х | х | х | Х | Х | х | Х | х | х | х | х | х | х |
| Age | < 40 | X | X | Х | X | X | X | X | х | X | X | х | X | Х | X | Х | Х | х | X |
| | 40-64 | Х | х | х | Х | х | Х | х | х | х | X | х | X | х | Х | х | х | х | х |
| | >=65 | х | х | х | x | х | х | х | х | х | X | х | X | х | х | х | х | х | х |
| Baseline Clinical Status | 7 | х | х | х | X | х | Х | х | х | х | Х | х | Х | х | х | х | х | х | х |
| | 6 | X | х | х | X | х | Х | х | х | х | X | х | Х | х | х | х | х | х | х |
| | continue for other scores | Х | х | х | Х | х | Х | Х | х | х | Х | х | X | х | Х | х | х | х | Х |

| | | | В | aricitini | b + RD | V | | | 1 | Placebo | + RDV | 7 | | | | All Su | bjects | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | erate<br>=X) | | /ere<br>=X) | 1 | bjects<br>=X) | | erate<br>=X) | 1 | vere<br>=X) | | bjects<br>=X) | | erate<br>=X) | | ere<br>=X) | | ubjects<br>=X) |
| Demographic Category | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Duration of Symptoms | Categorization 1 | X | х | х | х | х | Х | X | Х | х | X | х | Х | X | X | Х | Х | х | Х |
| prior to enrollment | Continue for all symptom categorizations | х | X | х | х | х | х | х | x | х | х | х | х | х | Х | х | х | х | х |
| Comorbidities | Comorbidity 1 | X | X | х | х | х | х | X | Х | х | Х | x | х | X | X | х | х | х | х |
| | Comorbidity 2 | X | X | Х | Х | х | Х | X | Х | х | Х | х | Х | X | Х | Х | X | Х | Х |
| | Continue for all comorbidities | х | х | х | х | х | х | х | х | х | х | x | х | х | Х | х | х | х | х |
| Comorbidities Group X | Continue for all comorbidity categorizations | x | x | х | х | x | x | х | х | х | x | x | x | x | х | x | x | х | x |

Table 51: Continuous Demographic and Baseline Characteristics by Randomized Disease Severity and Treatment Group – ITT Population

| | | E | Saricitinib + RE | V | | Placebo + RDV | • | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Statistic | Moderate<br>(N=X) | Severe<br>(N=X) | All Subjects<br>(N=X) | Moderate<br>(N=X) | Severe<br>(N=X) | All Subjects<br>(N=X) | Moderate<br>(N=X) | Severe<br>(N=X) | All Subjects<br>(N=X) |
| Age (years) | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | IQR | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | X | Х | х | X | Х | X | X | Х | X |
| | Maximum | X | Х | Х | X | Х | X | X | Х | X |
| Height (cm) | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | IQR | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | X | X | X | X | Х | X | X | X | X |
| | Maximum | X | X | X | X | Х | X | X | X | X |
| Weight (Kg) | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | IQR | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | X | X | X | X | Х | X | X | X | X |
| | Maximum | X | X | X | X | Х | X | X | X | X |
| BMI | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | IQR | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| | Minimum | X | X | X | X | X | X | X | X | X |
| | Maximum | X | X | x | X | х | x | X | x | X |

| | | В | Saricitinib + RD | V | | Placebo + RDV | | All Subjects | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Statistic | Moderate<br>(N=X) | Severe<br>(N=X) | All Subjects (N=X) | Moderate<br>(N=X) | Severe<br>(N=X) | All Subjects (N=X) | Moderate<br>(N=X) | Severe<br>(N=X) | All Subjects<br>(N=X) |
| Duration of Symptoms<br>prior to Enrollment (Days) | Mean | x.x | X.X | x.x | x.x | x.x | x.x | x.x | x.x | x.x |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | IQR | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | Х | X | X | Х | X | X | Х | X | X |
| | Maximum | Х | X | X | X | Х | х | X | X | X |

IQR is the inter-quartile range.

Table 52: Summary of Subjects with Pre-Existing Medical Conditions Treatment Group - As Treated Population

| | Baricitini<br>(N= | | Placebo<br>(N= | + RDV<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|
| Condition | n | % | n | % | n | % |
| None | X | XX | x | XX | Х | XX |
| Any Condition | X | XX | x | XX | Х | XX |
| Diabetes I | Х | XX | X | XX | Х | XX |
| Diabetes II | х | XX | X | XX | Х | XX |
| continue for all solicited conditions | | | | | | |

N = Number of subjects in the As Treated Population;

Programming Note: "None" and "Any Condition" will be the first two rows. The remainder of the rows will be sorted in order of prevalence, with the condition most reported among All Subjects being displayed first.

n = Number of subjects reporting the condition. Subjects who report 'unknown' for a condition are assumed to not have the condition.

Table 53: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification, Actual Disease Severity, and Treatment Group – As Treated Population

| | | | | ib + RDV<br>=X) | | | | + RDV<br>=X) | | | | ibjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic | WHO Drug Code<br>Level 2, Therapeutic | | erate<br>=X) | | vere<br>=X) | | erate<br>=X) | | vere<br>=X) | | erate<br>=X) | | vere<br>=X) |
| Group | Subgroup | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | Х | xx | x | xx | X | XX | X | XX | X | XX | X | XX |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | Х | xx | х | xx | x | XX | X | XX | X | xx | х | XX |
| | [ATC 2 - 1] | Х | xx | х | xx | x | XX | X | XX | X | xx | х | XX |
| | [ATC 2 - 2] | X | xx | x | xx | x | XX | X | XX | X | xx | х | XX |
| | [ATC 2 - 3] | X | xx | х | xx | x | XX | X | XX | X | xx | х | XX |
| [ATC Level 1 – 2] | [ATC 2 - 1] | X | xx | х | xx | x | XX | X | XX | X | xx | х | XX |
| | [ATC 2 - 2] | X | xx | x | xx | X | XX | X | XX | X | xx | x | xx |
| | [ATC 2 - 3] | Х | xx | х | xx | X | XX | X | XX | X | xx | x | xx |

N = Number of subjects in the As Treated Population.

n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

Programming Note: Only include medications with missing end dates (i.e. ongoing) or end dates on or after the enrollment date.

Table 54: Number and Percentage of Subjects Reporting Use of Medications of Interest by Actual Disease Severity, and Treatment Group – As Treated Population

| | | | inib + RDV<br>N=X) | | | | + RDV<br>=X) | | | | ıbjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | oderate<br>N=X) | | vere<br>=X) | | lerate<br>(=X) | | vere<br>=X) | | erate<br>=X) | | vere<br>=X) |
| Medication/Therapies | N | % | n | % | n | % | n | % | n | % | n | % |
| Any Medication/Therapy | Х | XX | х | xx | х | xx | х | xx | х | xx | х | xx |
| Protease inhibitors | X | XX | X | xx | Х | xx | х | xx | х | xx | х | xx |
| Polymerase inhibitors | X | XX | X | xx | Х | xx | х | xx | х | xx | х | xx |
| Potential Treatments for COVID-19 | X | XX | х | xx | Х | xx | х | xx | х | xx | х | xx |
| Chloroquine/Hydroxychloroquine | X | XX | X | xx | Х | xx | х | xx | х | xx | х | xx |
| Other | X | XX | х | xx | Х | xx | х | xx | х | xx | х | xx |
| Corticosteroids | X | XX | х | xx | X | xx | X | xx | X | xx | Х | XX |
| Other anti-inflammatory drugs | Х | XX | х | xx | Х | xx | X | xx | X | xx | х | xx |
| Monoclonal Antibodies Targeting<br>Cytokines | X | XX | x | XX | x | XX | x | xx | X | xx | x | xx |
| Other Biologic Therapies | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |

N = Number of subjects in the As Treated Population.

Programming Note: only include medications where the end date is missing (i.e. ongoing) or end date is on or after enrollment date

n=Number of subjects reporting taking at least one medication in the specified category.

Table 55: Use of Medications of Interest by Study Day, Actual Disease Severity, and Treatment Group – As Treated Population

| | | Baricitini<br>(N= | ib + RDV<br>=X) | | | Placebo + RDV All Subjects (N=X) (N=X) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | lerate<br>=X) | Sev<br>(N= | rere<br>=X) | | lerate<br>=X) | Sev<br>(N= | vere<br>=X) | | lerate<br>=X) | Severe<br>(N=X) | |
| Study Day | n | % | n | % | n | % | n | % | n | % | n | % |
| | | | | | Any Med | ication of Inter | est | | | | | |
| Day 1 | X | Xx | X | XX | X | XX | X | XX | X | XX | X | XX |
| Day 3 | X | Xx | X | XX | X | xx | X | XX | X | xx | X | XX |
| Day 5 | X | Xx | X | XX | X | xx | X | XX | X | xx | X | XX |
| Day 8 | X | Xx | X | XX | X | xx | X | XX | X | xx | X | XX |
| Day 11 | X | Xx | X | XX | X | xx | X | XX | X | xx | X | XX |

<sup>...</sup>Repeat for all categories and sub-categories of the medications in Section 6.4

Programming Note: If the start date of the prohibited medication is on or before the specified (actual) study day, then the subject will be denoted as taking the med for that Study Day.

N = Number of subjects in the As Treated Population.

n=Number of subjects reporting taking at least one prohibited medication by the specified study day.

**Table 56:** Overall Summary of Adverse Events – As Treated Population

| | | F | Baricitini<br>(N= | | OV | | | | | o + RDV<br>=X) | V | | | | | ubjects<br>=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mode<br>(N=) | | Seve<br>(N= | | | everity<br>=X) | | erate<br>=X) | | vere<br>=X) | | Severity<br>I=X) | Mode<br>(N= | | | ere<br>=X) | Any Se<br>(N= | |
| Subjects <sup>a</sup> with | N | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one adverse event | X | X | х | X | x | X | X | х | X | Х | X | Х | X | х | X | X | х | X |
| At least one Severe or Life-threatening (Grade 3 or 4) adverse event | X | Х | х | Х | X | Х | X | Х | Х | Х | Х | X | X | Х | Х | х | х | X |
| At least one related adverse event | X | X | х | X | х | x | x | х | X | Х | X | X | x | Х | х | X | х | X |
| Moderate (Grade 2) | X | X | х | X | X | X | X | X | Х | X | X | X | X | х | X | X | х | X |
| Severe (Grade 3) | X | X | х | Х | х | X | X | х | X | X | X | х | х | X | Х | Х | х | X |
| Life-threatening (Grade 4) | X | Х | х | х | Х | X | X | Х | Х | X | X | X | X | х | х | Х | x | X |
| Severe or Life-Threatening (Grade 3 or 4) | X | X | х | Х | X | X | X | Х | X | X | X | X | X | Х | Х | Х | х | X |
| Death (Grade 5) | X | X | X | X | X | Х | X | Х | X | X | X | X | X | Х | Х | X | Х | X |
| At least one not related adverse event | X | X | х | X | х | х | X | х | X | X | X | Х | Х | х | х | х | х | X |
| Moderate (Grade 2) | X | X | X | Х | Х | X | X | Х | Х | X | X | X | X | Х | Х | Х | X | X |
| Severe (Grade 3) | X | X | X | Х | Х | X | X | Х | Х | X | X | X | X | Х | Х | Х | X | X |
| Life-threatening (Grade 4) | X | X | х | X | X | X | X | X | Х | X | X | X | X | х | X | X | х | X |
| Death (Grade 5) | X | X | X | X | Х | Х | Х | Х | X | X | Х | X | Х | Х | Х | Х | Х | X |
| At least one serious adverse event | X | X | х | Х | x | X | Х | x | Х | X | x | Х | Х | x | x | x | х | X |
| At least one serious adverse event with fatal outcome | X | х | Х | X | х | х | х | х | x | х | х | х | х | х | х | х | Х | X |
| At least one related serious adverse event | X | х | х | Х | X | X | X | Х | Х | X | X | X | X | Х | Х | Х | x | X |
| At least one related serious adverse event with fatal outcome | X | Х | Х | X | Х | X | X | Х | Х | Х | Х | X | X | х | х | х | Х | X |
| At least one adverse event leading to study drug discontinuation | X | х | Х | X | Х | Х | Х | Х | х | х | х | X | X | х | Х | Х | Х | X |
| At least one related adverse event leading to study drug discontinuation | X | х | Х | X | Х | Х | X | Х | х | х | Х | X | Х | х | Х | Х | Х | X |

| | | F | Baricitinil<br>(N= | | OV | | | ] | Placebo<br>(N= | + RDV<br>=X) | V | | | | | ubjects<br>=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Moder<br>(N=X | | | | Any Severity Moders (N=X) (N=X) | | | | ere<br>=X) | | Any Severity (N=X) | | erate<br>X) | Severe<br>(N=X) | | Any Sev<br>(N=2 | | |
| Subjects <sup>a</sup> with | N | % 1 | | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one adverse event leading to early termination <sup>b</sup> | X | X | х | X | X | Х | X | х | х | х | х | Х | X | Х | х | х | Х | X |
| At least one Unanticipated Problem | X | X X | | Х | Х | х | X | Х | X | X | Х | Х | X | Х | X | Х | X | X |

N = Number of subjects in the actual disease severity stratum and As Treated Population aSubjects are counted once for each category regardless of the number of events. bAs reported on the Adverse Event eCRF.

Programming Note: Use actual severity

All Grade 3 and 4 AEs are captured as AEs. In addition, any Grade 2 or higher suspected drug-related hypersensitivity reaction is reported as an AE.

Table 57: Subject-Level Rates of Adverse Events and Differences between Treatment Groups – As Treated Population

| | | nib + RDV<br>[=X] | | + RDV<br>=X) | |
|---|---|---|---|---|---|
| Subjects <sup>a</sup> with at least one: | n | % | n | % | Risk Difference (95% CI) |
| AE | X | Х | Х | х | x.x (x.x, x.x) |
| Related AE | X | Х | Х | х | x.x (x.x, x.x) |
| Grade 3-4 AE | X | Х | Х | х | x.x (x.x, x.x) |
| Grade 3-4 Related AE | X | Х | Х | х | x.x (x.x, x.x) |
| SAE | X | Х | Х | х | x.x (x.x, x.x) |
| Related SAE | X | Х | Х | х | x.x (x.x, x.x) |
| SAE with fatal outcome | X | Х | Х | х | x.x (x.x, x.x) |
| Related SAE with fatal outcome | X | Х | Х | х | x.x (x.x, x.x) |
| AE leading to discontinuation of study drug | X | Х | Х | х | x.x (x.x, x.x) |
| Related AE leading to discontinuation of study drug | X | х | х | х | x.x (x.x, x.x) |

N = Number of subjects in the As Treated Population.

<sup>&</sup>lt;sup>a</sup>Subjects are counted once for each category regardless of the number of events.

Table 58: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - As Treated Population

| Preferred Term | MedDRA System<br>Organ Class | Bar | icitinib<br>(N=X | | Pla | cebo + R<br>(N=X) | RDV | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events |
| PT1 | SOC1 | X | X | X | X | X | X | X | X | X |
| Etc. | Etc. | X | X | Х | X | X | Х | X | X | Х |

N = number of subjects in the As Treated Population (number of subjects at risk).

## **Programming Notes:**

Select all preferred terms/System organ classes where the % for any treatment group or overall is  $\ge 5\%$ . Sort preferred terms by descending order of frequency.

#### Tables with similar format:

Table 59: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA

System Organ Class and Preferred Term, and Treatment Group - Moderate Disease

**Severity, As Treated Population** 

Table 60: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA

System Organ Class and Preferred Term, and Treatment Group – Severe Disease

**Severity, As Treated Population** 

Programming Notes for Tables 59 and 60: Actual disease severity will be used.

n = number of subjects reporting event.

Events = total frequency of events reported.

**Table 61:** Treatment-Emergent Renal Adverse Events by Preferred Term and Treatment Group – As Treated Population

| Preferred Term | Baı | ricitinib +<br>(N=X) | RDV | Pl | acebo + R<br>(N=X) | DV | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|
| | n | % | Events | n | % | Events | n | % | Events |
| Any treatment-emergent hepatic adverse event | х | х | х | X | Х | х | X | х | X |
| Glomerular filtration rate decreased | x | Х | х | x | X | х | x | х | х |
| Blood creatinine increased | x | х | x | X | x | x | x | х | x |
| Acute kidney injury | x | х | x | X | x | x | x | х | x |
| Creatinine renal clearance decreased | x | х | X | x | x | x | x | х | х |
| Renal failure | x | х | x | X | x | x | x | х | x |
| Renal impairment | x | х | x | X | x | x | x | х | x |
| Proteinuria | x | х | x | X | x | x | x | х | x |
| Renal tubular necrosis | x | х | X | x | x | x | x | х | х |
| Blood creatinine abnormal | х | x | x | x | x | x | x | х | х |
| Continuous haemodiafiltration | x | Х | X | x | X | x | x | Х | х |
| Glomerular filtration rate abnormal | х | x | х | x | x | х | x | х | х |

N = Number of subjects in the As Treated Population.

Treatment-Emergent Hepatic Adverse Events by Preferred Term and Treatment Group **Table 62:** 

- As Treated Population

**Table 63:** Related Adverse Events by MedDRA System Organ Class and Preferred Term, and **Treatment Group - As Treated Population** 

| | | Bar | ricitinib<br>(N=X | | Pla | cebo + F<br>(N=X) | RDV | All Subjects (N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | Preferred Term | n | % | Events | n | % | Events | n | % | Events |
| Any SOC | Any PT | X | X | X | X | X | X | X | X | X |
| SOC1 | Any PT | X | X | X | X | X | X | X | X | X |
| Etc. | Etc. | | | | | | | | | |

N = number of subjects in the As Treated Population (number of subjects at risk).

n = Number of subjects reporting event.

Events = Total frequency of events reported.

n = number of subjects reporting event.

Events = total frequency of events reported.

Table 64: Deaths by Day 15 or Day 29 by Treatment Group and Randomized Disease Severity – ITT Population

| | Randomized Disease | | Baricitinib + RDV<br>(N=X) | | | Placebo + RDV<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Study Day | Severity | n | Mortality Rate <sup>a</sup> | Rate 95% CI | n | Mortality Rate <sup>a</sup> | Rate 95% CI |
| Day 15 | Moderate | X | X.X | x.x, x.x | X | x.x | X.X, X.X |
| | Severe | X | X.X | x.x, x.x | X | X.X | X.X, X.X |
| | Any Severity | X | X.X | x.x, x.x | X | X.X | X.X, X.X |
| Day 29 | Moderate | X | X.X | x.x, x.x | X | X.X | X.X, X.X |
| | Severe | X | x.x | x.x, x.x | X | x.x | x.x, x.x |
| | Any Severity | X | X.X | x.x, x.x | X | x.x | X.X, X.X |

N = Number of Subject in the specified treatment group and analysis population.

Table 65: Deaths by Day 15 or Day 29 by Treatment Group and Actual Disease Severity – As Treated Population

n = Number of subjects in a given treatment group who died by the given timepoint

<sup>&</sup>lt;sup>a</sup> Mortality Rate is the Kaplan-Meier estimate.

Table 66: Time to Death through Day 15 and 29 by Treatment Group and Randomized Disease Severity – ITT Population

| | | | | Media | an Time | Н | ₹ | |
|---|---|---|---|---|---|---|---|---|
| Study Day | Treatment Group | Randomized Disease Severity | n | Estimate | 95% CI | Estimate | 95% CI | P-value |
| Day 15 | Baricitinib + RDV (N=X) | Moderate | X | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | | X | x.x | x.x, x.x | x.xx | x.xx, x.xx | |
| | Baricitinib + RDV (N=X) | Severe | X | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | | X | x.x | x.x, x.x | x.xx | x.xx, x.xx | |
| | Baricitinib + RDV (N=X) | Any Severity | X | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | | X | x.x | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |
| Day 29 | Baricitinib + RDV (N=X) | Moderate | Х | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | | X | x.x | x.x, x.x | x.xx | x.xx, x.xx | |
| | Baricitinib + RDV (N=X) | Severe | X | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | | X | x.x | x.x, x.x | x.xx | x.xx, x.xx | |
| | Baricitinib + RDV (N=X) | Any Severity | X | x.x | x.x, x.x | | | |
| _ | Placebo + RDV (N=X) | | Х | X.X | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |

N= Number of subjects in the specified treatment group and analysis population.

Table 67: Time to Death through Day 15 and 29 by Treatment Group and Actual Disease Severity – As Treated Population

Table 68: Time to Death through Day 15 and 29 by Treatment Group within Subgroups – ITT Population

Table 69: Time to Death through Day 15 and 29 by Treatment Group: Medications of Interest Sensitivity Analysis – ITT Population

Table 70: Time to Death through Day 15 and 29 by Treatment Group: Interaction Modeling – ITT Population

# Programming notes for Table 68:

Log-rank p-values will not be included in this table so the column will be removed. The Disease Severity column will be removed and to the left of the Study Day column, a column titled "Analysis/Subgroup" will be inserted. Rows will be generated for each subgroup.

n = Number of subjects who died by the specified study day.

HR is the ratio of the hazard of Death in each treatment group estimated from the stratified Cox model. The ratio is Baricitinib + RDV to Placebo + RDV.

P-value calculated using the stratified Log-rank test.

# Programming notes for Table 69:

Log-rank p-values will not be included in this table so the column will be removed. The table will include a column to the left of the "n" column titled "m". The corresponding footnote will read "m = Number of subjects reporting use of the medication of interest." The Disease Severity column will be removed and a "Medication of Interest" column will be inserted to the left of Study Day. Separate models will be fit for the following categories of medications (see Section 6.4):

- Any Medication of Interest
- Hydroxychloroquine/Chloroquine
- Corticosteroids
- Anti-Inflammatory Drugs

The table will include the following footnote: "In this analysis, subjects that reported use of the specified medications of interest (Section 6.4 of the SAP) are censored at time of medication receipt."

## Programming notes for Table 70:

This table will only include the Treatment Group and HR columns only as well as a column to the left of Treatment Group titled "Interaction". Two models will be run: "Treatment – Randomized Disease Severity" will include a treatment\*randomized disease severity interaction term. "Treatment – Baseline Ordinal Score" will include a treatment\*baseline ordinal score interaction term. For each interaction model, the p-value for the interaction term will be provided in a footnote reading "The p-value for the treatment by [randomized disease severity/baseline ordinal score] interaction term was 0.xxxx.".

Time to Death through Day 15 and 29 by Treatment Group: Restricted Mean Survival Time Analysis – ITT Population **Table 71:** 

| | | | | Restricted Mea | nn Recovery Time | Differ | ence |
|---|---|---|---|---|---|---|---|
| Study Day | Treatment Group | Randomized Disease Severity | n | Estimate | 95% CI | Estimate | 95% CI |
| Day 15 | Baricitinib + RDV (N=X) | 36.1 | Х | x.x | x.x, x.x | | |
| | Placebo + RDV (N=X) | Moderate | X | X.X | x.x, x.x | X.XX | x.xx, x.xx |
| | Baricitinib + RDV (N=X) | G | Х | X.X | x.x, x.x | | |
| | Placebo + RDV (N=X) | Severe | Х | x.x | x.x, x.x | X.XX | x.xx, x.xx |
| | Baricitinib + RDV (N=X) | | Х | x.x | x.x, x.x | | |
| | Placebo + RDV (N=X) | Any Severity | Х | X.X | x.x, x.x | X.XX | x.xx, x.xx |
| Day 29 | Baricitinib + RDV (N=X) | M. J | Х | X.X | x.x, x.x | | |
| | Placebo + RDV (N=X) | Moderate | Х | X.X | x.x, x.x | X.XX | X.XX, X.XX |
| | Baricitinib + RDV (N=X) | G | Х | X.X | x.x, x.x | | |
| | Placebo + RDV (N=X) | Severe | Х | X.X | x.x, x.x | X.XX | x.xx, x.xx |
| | Baricitinib + RDV (N=X) Placebo + RDV (N=X) | Any Severity | Х | X.X | x.x, x.x | | |
| | | | Х | x.x | x.x, x.x | X.XX | x.xx, x.xx |

N= Number of subjects in the specified treatment group, disease severity, and analysis population. n= Number of subjects who died by the specified study day.

Difference is the difference in the restricted mean mortality time between Baricitinib + RDV and Placebo + RDV.

Table 72: Subjects Experiencing Grade 3 or 4 AEs and SAEs through Day 29 by Treatment Group and Actual Disease Severity – As Treated Population

| | | Baricitinib + RDV | | | Placebo + RDV | | |
|---|---|---|---|---|---|---|---|
| Safety Event Outcome | n | % | 95% CI | n | % | 95% CI | P-value |
| | | | Any Severity (N = 2 | K) | | | |
| Grade 3 or 4 AE | X | X | x.x, x.x | X | X | x.x, x.x | 0.xxx |
| SAE | X | X | x.x, x.x | X | X | x.x, x.x | 0.xxx |
| | | | Moderate (N = X) | | | | |
| Grade 3 or 4 AE | X | X | x.x, x.x | Х | X | x.x, x.x | 0.xxx |
| SAE | X | X | x.x, x.x | Х | X | x.x, x.x | 0.xxx |
| | | | Severe (N = X) | | | | |
| Grade 3 or 4 AE | X | X | x.x, x.x | Х | X | x.x, x.x | 0.xxx |
| SAE | X | X | x.x, x.x | Х | X | x.x, x.x | 0.xxx |

N = Number of Subject in the As Treated Population and specified actual disease severity stratum.

n = Number of subjects in a given treatment group who experienced the specified safety event outcome.

<sup>95%</sup> CI calculated using C-P/Blaker method

P-value calculated using Barnard's Exact Test

Table 73: Analysis of Time to Death, SAEs, or Grade 3 or 4 AEs by Treatment Group – As Treated Population

| | | | Medi | an Time | Н | <u> </u> | P-value |
|---|---|---|---|---|---|---|---|
| Actual Disease Severity | Treatment Group | n | Estimate | 95% CI | Estimate | 95% CI | |
| Any Severity (N=X) | Baricitinib + RDV (N=X) | X | x.x | x.x, x.x | | | |
| | Placebo + RDV (N=X) | X | X.X | x.x, x.x | x.xx | x.xx, x.xx | x.xxx |
| Moderate (N=X) | Baricitinib + RDV (N=X) | X | X.X | x.x, x.x | | | |
| | Placebo + RDV (N=X) | X | X.X | x.x, x.x | x.xx | x.xx, x.xx | |
| Severe (N=X) | Baricitinib + RDV (N=X) | X | X.X | x.x, x.x | | | |
| | Placebo + RDV (N=X) | X | X.X | x.x, x.x | x.xx | x.xx, x.xx | |

N= Number of subjects in the As Treated Population and specified actual disease severity stratum.

n = Number of subjects who died or experienced SAEs or Grade 3 or 4 AEs.

HR is the ratio of the hazard of Death/SAE/AE of Grade 3 or 4 in each treatment group estimated from the stratified Cox model. The ratio is Baricitinib + RDV to Placebo + RDV.P-value calculated using the Log-rank test

Table 74: Infections by Treatment Group – As Treated Population, Moderate Disease Severity

| | | | | | Bari | citinib +<br>(N=X) | RDV | | | | | | | | ebo + Rl<br>(N=X) | OV | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Anatomical | | | Sevei | re | Life | -Threate | ning | | Deatl | 1 | | Sever | e | Life- | Threate | ning | | Death | 1 |
| Location | Pathogen | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Any Location | Any Pathogen | х | х | x | Х | х | X | X | Х | Х | х | х | Х | х | х | X | Х | х | х |
| | Any Pathogen | X | X | X | X | X | X | x | X | х | x | х | X | X | х | х | x | х | x |
| Location 1 | Pathogen 1 | х | х | х | х | х | X | X | х | Х | х | х | х | Х | х | х | Х | х | х |
| | Pathogen 2 | х | х | х | Х | х | X | X | х | X | X | х | х | Х | х | х | Х | х | х |
| | Any Pathogen | х | х | X | X | х | X | X | х | Х | Х | х | X | x | х | X | Х | х | Х |
| Location 2 | Pathogen 1 | х | х | X | X | х | X | X | X | Х | Х | х | х | x | Х | X | Х | х | X |
| | Pathogen 2 | X | X | X | x | x | X | X | X | Х | Х | х | X | X | х | X | X | х | X |

Note: Percents may not add to 100 because participants may have infections with multiple pathogens. All Grade 3 or 4 infections are also reported as AEs.

N=Number of participants randomized to Treatment group.

n=Number of participants with infection.

#### Tables with similar format:

Table 75: Opportunistic Infections by Treatment Group – As Treated Population, Moderate Disease Severity

Table 76: Infections by Treatment Group – As Treated Population, Severe Disease Severity

Table 77: Opportunistic Infections by Treatment Group – As Treated Population, Severe Disease Severity

Table 78: Infections by Treatment Group – As Treated Population, All Subjects

Table 79: Opportunistic Infections by Treatment Group – As Treated Population, All Subjects

Programming Notes for Table 75, Table 77, Table 79: Opportunistic infections will be identified by the sponsor and will be documented in a spreadsheet/SAS dataset to be imported into ADaM dataset programming.

Table 80: Abnormal Laboratory Results of Grade 3 or 4 by Parameter, Maximum Severity, Time Point, and Treatment Group – As Treated Population

| Laboratory | | | | Severe/ | Grade 3 | Life Threate | ning/ Grade 4 | | brade 3 or<br>ning/Grade 4 |
|---|---|---|---|---|---|---|---|---|---|
| Parameter Parameter | Time Point | Treatment Group | N | n | % | n | % | n | % |
| Any Parameter | Baseline | Baricitinib + RDV | X | x | х | X | X | X | X |
| | | Placebo + RDV | X | x | X | X | X | X | X |
| | Day 3 | Baricitinib + RDV | X | X | X | х | Х | x | X |
| | | Placebo + RDV | X | х | X | х | Х | x | X |
| | Day 5 | Baricitinib + RDV | X | х | X | х | Х | x | X |
| | | Placebo + RDV | x | х | X | х | Х | х | X |
| | Day 8 | Baricitinib + RDV | x | х | X | х | Х | х | X |
| | | Placebo + RDV | x | х | X | х | Х | х | x |
| | Day 11 | Baricitinib + RDV | X | х | X | х | Х | x | X |
| | | Placebo + RDV | x | х | X | х | Х | х | X |
| | Day 15 | Baricitinib + RDV | x | х | X | х | Х | х | X |
| | | Placebo + RDV | x | х | X | х | Х | х | X |
| | Day 29 | Baricitinib + RDV | x | х | X | х | Х | х | X |
| | | Placebo + RDV | x | х | X | х | х | х | х |
| | Maximum Severity Post<br>Baseline | Baricitinib + RDV | Х | x | X | X | х | x | х |
| | | Placebo + RDV | Х | X | X | X | Х | X | X |

Each parameter will be summarized individually similar to the above...

The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments and assessments beyond Day 29.

N = Number of subjects in the As Treated Population

Programming Note: D-dimer and CRP results are not included in this table. Include all lab parameters that are being graded in this table.

- Table 81: Abnormal Laboratory Results of Grade 3 or 4 by Parameter, Maximum Severity, Time Point, and Treatment Group Moderate Disease Severity, As Treated Population
- Table 82: Abnormal Laboratory Results of Grade 3 or 4 by Parameter, Maximum Severity, Time Point, and Treatment Group Severe Disease Severity, As Treated Population

Programming Notes for Table 81 and Table 82: Actual Disease Severity will be used. Include all lab parameters that are being graded in this table.

**Table 83:** Treatment-Emergent Laboratory Abnormalities - As Treated Population

| | | | Baricitinib + RI<br>(N=X) | OV | Placebo + RDV<br>(N=X) | | |
|---|---|---|---|---|---|---|---|
| <b>Laboratory Parameter</b> | Grade | N | n | % | N | n | % |
| Any Parameter | 1 | X | X | X | X | X | X |
| | 2 | X | Х | X | X | X | X |
| | 3 | X | Х | X | X | X | X |
| | 4 | х | Х | X | X | X | X |
| | Any Grade | X | Х | X | X | X | X |

Continue for all graded parameters

N = number of subjects in the As Treated Population with any post-baseline data available for the specified Lab Parameter.

n = number of subjects in the As Treated Population with treatment emergent abnormalities for the specified Lab Parameter.

A treatment emergent laboratory abnormality is defined as a post-baseline abnormal value with a severity grade greater than at baseline.

Table 84: Summary Statistics of Laboratory Results by Parameter, Study Visit Day, and Treatment Group – As Treated Population

| Laboratory | | | Absolute | | | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Parameter | Study Visit Day | Treatment Group | N | Mean | SD | Median | Min, Max | N | Mean | SD | Median | Min, Max |
| Parameter 1 | Baseline | Baricitinib + RDV | X | xx.x | XX.X | XX.X | xx.x, xx.x | | | | | |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | | | | | |
| | Day 3 | Baricitinib + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | Day 5 | Baricitinib + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | Day 8 | Baricitinib + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | Day 11 | Baricitinib + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | Day 15 | Baricitinib + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | xx.x | xx.x | xx.x, xx.x |
| | Day 29 | Baricitinib + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | xx.x | xx.x | xx.x, xx.x |
| | | Placebo + RDV | x | xx.x | xx.x | xx.x | xx.x, xx.x | X | XX.X | XX.X | xx.x | xx.x, xx.x |

Continue for all parameters...

N = Number of subjects in the As Treated Population with laboratory data available for the parameter at the specified study visit.

Programming Notes: Include all lab parameters in this table.

Tables with similar format:

Table 85: Summary Statistics of Laboratory Results by Parameter, Study Visit Day, and Treatment Group – Moderate Disease Severity, As Treated Population

Table 86: Summary Statistics of Laboratory Results by Parameter, Study Visit Day, and Treatment Group – Severe Disease Severity, As Treated Population

Programming Notes for Tables 85 and 86: Actual Disease Severity will be used. Include all lab parameters in this table.

## **APPENDIX 2. FIGURE MOCK-UPS**

General Programming Notes for figures:

- Treatment group labeling will be the following:
  - o Baricitinib + RDV
  - o Placebo + RDV
- If the treatment group labels need to be abbreviated to improve fit, the following abbreviations will be used:
  - $\circ$  B+R
  - $\circ$  P+R
- Use the same color for a treatment on the different graphs:
  - o Baricitinib + RDV = Blue
  - $\circ$  Placebo + RDV = Red
- For severity graphs:
  - $\circ$  Mild = yellow
  - Moderate = orange
  - Severe = light red
  - o Life-threatening = red
  - $\circ$  Death = black

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 106 |
|---|---|---|
| Figure 2: | Kaplan-Meier Curves of Time to Recovery by Treatment Group – ITT Population | 107 |
| Figure 3: | Kaplan-Meier Curve of Time to Recovery by Treatment Group – As Treated Population | 108 |
| Figure 4: | Kaplan-Meier Curve of Time to Recovery by Treatment Group and Randomized Disease Severity – ITT Population | 108 |
| Figure 5: | Kaplan-Meier Curve of Time to Recovery by Treatment Group and Randomized Disease Severity – As Treated Population | 108 |
| Figure 6: | Kaplan-Meier Curve of Time to Recovery by Treatment Group – Baseline Ordinal Score 7, ITT Population | 108 |
| Figure 7: | Kaplan-Meier Curve of Time to Recovery by Treatment Group – Baseline Ordinal Score 6, ITT Population | 108 |
| Figure 8: | Kaplan-Meier Curve of Time to Recovery by Treatment Group – Baseline Ordinal Score 5, ITT Population | 108 |
| Figure 9: | Kaplan-Meier Curve of Time to Recovery by Treatment Group – Baseline Ordinal Score 4, ITT Population | 108 |
| Figure 10: | Forest Plot of Hazard Ratios of Time to Recovery by Subgroup - ITT Population | 109 |
| Figure 11: | Forest Plot of Hazard Ratios of Time to Recovery by Subgroup - As Treated Population | 109 |
| Figure 12: | Forest Plot of Hazard Ratios of Time to Recovery by Comorbidity - ITT Population | 109 |
| Figure 13: | Forest Plot of Hazard Ratios of Time to Recovery: Leave One Site Out<br>Sensitivity Analysis - ITT Population | 109 |
| Figure 14: | Study Visit Day 15 Clinical Status Score by Baseline Score and Treatment Group – ITT Population | |
| Figure 15: | Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group – ITT Population | 111 |
| Figure 16: | Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group – ITT Population | |
| Figure 17: | Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group – Baseline Ordinal Score 7, ITT Population | |
| Figure 18: | Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group – Baseline Ordinal Score 6, ITT Population | 112 |

| Figure 19: | Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group – Baseline Ordinal Score 5, ITT Population | 112 |
|---|---|---|
| Figure 20: | Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group – Baseline Ordinal Score 4, ITT Population | 112 |
| Figure 21: | Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group – Baseline Ordinal Score 7, ITT Population | 112 |
| Figure 22: | Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group – Baseline Ordinal Score 6, ITT Population | 112 |
| Figure 23: | Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group – Baseline Ordinal Score 5, ITT Population | 112 |
| Figure 24: | Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group – Baseline Ordinal Score 4, ITT Population | 112 |
| Figure 25: | Distribution of Clinical Status Scores by Day by Treatment Group – ITT Population | 113 |
| Figure 26: | Bar Plots of Clinical Status Scores by Study Day and Treatment Group – ITT Population | 114 |
| Figure 27: | Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group – ITT Population | 115 |
| Figure 28: | Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group – Baseline Ordinal Score 7, ITT Population | 115 |
| Figure 29: | Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group – Baseline Ordinal Score 6, ITT Population | 115 |
| Figure 30: | Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group – Baseline Ordinal Score 5, ITT Population | 115 |
| Figure 31: | Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group – Baseline Ordinal Score 4, ITT Population | 115 |
| Figure 32: | Mean NEWS by Day and Treatment Group – ITT Population | 116 |
| Figure 33: | Bee Swarm Plot of Oxygen Days by Treatment Group – ITT Population | 117 |
| | Bee Swarm Plot of Non-invasive Ventilation/High-Flow Oxygen Days by Treatment Group – ITT Population | |
| Figure 35: | Bee Swarm Plot of Invasive Mechanical Ventilation/ECMO Days by Treatment Group – ITT Population | 117 |

| Figure 36: | Bee Swarm Plot of Hospitalization Days by Treatment Group – ITT Population | 117 |
|---|---|---|
| Figure 37: | Frequency of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group - As Treated Population | 118 |
| Figure 38: | Frequency of Non-Serious Related Adverse Events by MedDRA System<br>Organ Class, Severity, and Treatment Group – Moderate Disease Severity,<br>As Treated Population | 118 |
| Figure 39: | Frequency of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Severe Disease Severity, As Treated Population | 118 |
| Figure 40: | Incidence of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group - As Treated Population | 119 |
| Figure 41: | Incidence of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Moderate Disease Severity, As Treated Population | 119 |
| Figure 42: | Incidence of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Severe Disease Severity, As Treated Population | 119 |
| Figure 43: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group — ITT Population | 120 |
| Figure 44: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group and Randomized Disease Severity – ITT Population | 121 |
| Figure 45: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group – As Treated Population | 121 |
| Figure 46: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group and Actual Disease Severity – As Treated Population | 121 |
| Figure 47: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group – Baseline Ordinal Score 7, ITT Population | 121 |
| Figure 48: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group – Baseline Ordinal Score 6, ITT Population | 121 |
| Figure 49: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group – Baseline Ordinal Score 5, ITT Population | 121 |
| Figure 50: | Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group – Baseline Ordinal Score 4, ITT Population | 121 |
| Figure 51: | Kaplan-Meier Curve of Time to Death, SAE, Discontinuation of Study<br>Infusions or Grade 3 or 4 AE through Day 29 by Treatment Group – As<br>Treated Population | 122 |

| Statistical Analy | sis Plan - | <b>DMID</b> | Protocol: | 20-0006 | (ACTT-2) |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| Version | 3.0 |
|---------|-----|
| 0AUG2 | 020 |

| Figure 52: | Kaplan-Meier Curve of Time to Death, SAE, Discontinuation of Study<br>Infusions or Grade 3 or 4 AE through Day 29 by Treatment Group and<br>Actual Disease Severity – As Treated Population | 122 |
|---|---|---|
| Figure 53: | [Parameter X] Results by Scheduled Visits: Change from Baseline by Treatment Group – As Treated Population | 123 |

Figure 1: CONSORT Flow Diagram



Programming Note: Disease Stratum will be included in the final CONSORT diagram as separate diagrams. Content of individual boxes may be altered from the shell.



Figure 2: Kaplan-Meier Curves of Time to Recovery by Treatment Group – ITT Population

Programming Note: For Subjects at risk counts, only display Days 1, 3, 5, 8, 11, 15, 22, 29. Report p-value to 3 decimal places as noted in Section 13.

Figures with similar format:

- Figure 3: Kaplan-Meier Curve of Time to Recovery by Treatment Group As Treated Population
- Figure 4: Kaplan-Meier Curve of Time to Recovery by Treatment Group and Randomized Disease Severity ITT Population
- Figure 5: Kaplan-Meier Curve of Time to Recovery by Treatment Group and Randomized Disease Severity As Treated Population
- Figure 6: Kaplan-Meier Curve of Time to Recovery by Treatment Group Baseline Ordinal Score 7, ITT Population
- Figure 7: Kaplan-Meier Curve of Time to Recovery by Treatment Group Baseline Ordinal Score 6, ITT Population
- Figure 8: Kaplan-Meier Curve of Time to Recovery by Treatment Group Baseline Ordinal Score 5, ITT Population
- Figure 9: Kaplan-Meier Curve of Time to Recovery by Treatment Group Baseline Ordinal Score 4, ITT Population


Figure 10: Forest Plot of Hazard Ratios of Time to Recovery by Subgroup - ITT Population

Figures with similar format:

Figure 11: Forest Plot of Hazard Ratios of Time to Recovery by Subgroup - As Treated Population

Figure 12: Forest Plot of Hazard Ratios of Time to Recovery by Comorbidity - ITT Population

Figure 13: Forest Plot of Hazard Ratios of Time to Recovery: Leave One Site Out Sensitivity

**Analysis - ITT Population** 

Programming Notes for Figure 12: Use the comorbidities listed in Table 52.

Figure 14: Study Visit Day 15 Clinical Status Score by Baseline Score and Treatment Group – ITT Population



Figure 15: Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group – ITT Population



Figure with similar format:

- Figure 16: Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group ITT Population
- Figure 17: Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group Baseline Ordinal Score 7, ITT Population
- Figure 18: Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group Baseline Ordinal Score 6, ITT Population
- Figure 19: Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group Baseline Ordinal Score 5, ITT Population
- Figure 20: Kaplan-Meier Curves of Time to Improvement by at least One Category of Clinical Status Score by Treatment Group Baseline Ordinal Score 4, ITT Population
- Figure 21: Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group Baseline Ordinal Score 7, ITT Population
- Figure 22: Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group Baseline Ordinal Score 6, ITT Population
- Figure 23: Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group Baseline Ordinal Score 5, ITT Population
- Figure 24: Kaplan-Meier Curves of Time to Improvement by at least Two Categories of Clinical Status Score by Treatment Group Baseline Ordinal Score 4, ITT Population



Figure 25: Distribution of Clinical Status Scores by Day by Treatment Group – ITT Population

Programming Note: Heat map coloring will be used for the clinical score scale. The y-axis will be percentages instead of frequency counts. The same categories presented in the tabular summary will be use in this figure. The "no clinical score" categories will displayed at the top of the stacked bars using colors distinct from the heat map colors. Use the format/coloring used for ACTT-1.



Programming Note: The same categories presented in the tabular summary will be use in this figure. The "no clinical score" categories will be displayed at the x = 9, 10, 11 (and 12 if the Completed Study without reporting score category is needed).

Figure 27: Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group – ITT Population



Figures with similar format:

- Figure 28: Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group Baseline Ordinal Score 7, ITT Population
- Figure 29: Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group Baseline Ordinal Score 6, ITT Population
- Figure 30: Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group Baseline Ordinal Score 5, ITT Population
- Figure 31: Kaplan-Meier Curves of Time to Discharge or NEWS ≤ 2 by Treatment Group Baseline Ordinal Score 4, ITT Population



Figure 32: Mean NEWS by Day and Treatment Group – ITT Population

Programming Note: Add the footnote: Subjects who die or are discharged are not reflected in Study Days after their date of death/discharge.



Figure 33: Bee Swarm Plot of Oxygen Days by Treatment Group – ITT Population

Programming Note: Use the format used for ACTT-1 which incorporated summary statistics.

Figures with similar format:

- Figure 34: Bee Swarm Plot of Non-invasive Ventilation/High-Flow Oxygen Days by Treatment Group ITT Population
- Figure 35: Bee Swarm Plot of Invasive Mechanical Ventilation/ECMO Days by Treatment Group ITT Population
- Figure 36: Bee Swarm Plot of Hospitalization Days by Treatment Group ITT Population

Figure 37: Frequency of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group - As Treated Population



Programming Note: Two separate sub-figures will be generated for each disease severity. Actual disease severity will be used for each figure.

#### Figures with similar format:

Figure 38: Frequency of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Moderate Disease Severity, As Treated Population

Figure 39: Frequency of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Severe Disease Severity, As Treated Population

Figure 40: Incidence of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group - As Treated Population



Programming Note: Two separate sub-figures will be generated for each disease severity. Actual disease severity will be used for each figure.

#### Figures with similar format:

Figure 41: Incidence of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Moderate Disease Severity, As Treated Population

Figure 42: Incidence of Non-Serious Related Adverse Events by MedDRA System Organ Class, Severity, and Treatment Group – Severe Disease Severity, As Treated Population

Figure 43: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group – ITT Population



Figures with similar format:

- Figure 44: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group and Randomized Disease Severity ITT Population
- Figure 45: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group As Treated Population
- Figure 46: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group and Actual Disease Severity As Treated Population
- Figure 47: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group Baseline Ordinal Score 7, ITT Population
- Figure 48: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group Baseline Ordinal Score 6, ITT Population
- Figure 49: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group Baseline Ordinal Score 5, ITT Population
- Figure 50: Kaplan-Meier Curve of Time to Death through Day 29 by Treatment Group Baseline Ordinal Score 4, ITT Population

Programming Notes for Figure 44 and Figure 46: The figures will have two panels, one for each disease severity.

Figure 51: Kaplan-Meier Curve of Time to Death, SAE, Discontinuation of Study Infusions or Grade 3 or 4 AE through Day 29 by Treatment Group – As Treated Population



Figure with similar format:

Figure 52: Kaplan-Meier Curve of Time to Death, SAE, Discontinuation of Study Infusions or Grade 3 or 4 AE through Day 29 by Treatment Group and Actual Disease Severity – As Treated Population

Programming Note: Figure will have two panels, one for each disease severity.

Figure 53: [Parameter X] Results by Scheduled Visits: Change from Baseline by Treatment Group – As Treated Population



Programming Note: The shell provided is a generic figure. The Groups within a panel will be treatment groups and the panels will be actual disease severity. The points will be the median change from baseline and the bars will represent the Q1 and Q3 quartiles of the change from baseline at each time point. Panels for each laboratory parameter will be generated.

## APPENDIX 3. LISTINGS MOCK-UPS

## **TABLE OF LISTINGS**

| Listing 1: | Exclusions from the As Treated Population | 125 |
|---|---|---|
| Listing 2: | Subjects who Early Terminated or Discontinued Treatment | 126 |
| Listing 3: | Subject-Specific Protocol Deviations | 127 |
| Listing 4: | Non-Subject-Specific Protocol Deviations | 128 |
| Listing 5: | Individual Efficacy Response Data: Clinical Status Score Data | 129 |
| Listing 6: | Individual Efficacy Response Data: NEWS | 130 |
| Listing 7: | Demographic Data | 131 |
| Listing 8: | Pre-Existing and Concurrent Medical Conditions | 132 |
| Listing 9: | Concomitant Medications | 133 |
| Listing 10: | Medications of Interest | 134 |
| Listing 11: | Compliance Data | 135 |
| Listing 12: | Listing of Non-Serious Adverse Events | 136 |
| Listing 13: | Listing of Related Adverse Events | 137 |
| Listing 14: | Listing of Non-Fatal Serious Adverse Events | 138 |
| Listing 15: | Listing of Infections | 139 |
| Listing 16: | Listing of Deaths | 140 |
| Listing 17: | Pregnancy Reports – Maternal Information | 141 |
| Listing 18: | Pregnancy Reports – Gravida and Para | 142 |
| Listing 19: | Pregnancy Reports – Live Birth Outcomes | 143 |
| Listing 20: | Pregnancy Reports – Still Birth Outcomes | 144 |
| Listing 21: | Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 145 |
| Listing 22: | Clinical Laboratory Results | 146 |
| Listing 23: | Physical Exam Findings | 147 |
| Listing 24: | Subjects who Received the Incorrect Treatment | 148 |
| Listing 25: | Subjects Randomized to the Incorrect Disease Severity Stratum | 148 |

**Listing 1:** Exclusions from the As Treated Population

| Randomized Treatment Group | Actual Disease Severity | Subject ID |
|----------------------------|-------------------------|------------|
| Baricitinib + RDV/ | Moderate / Severe | XXXXX |
| Placebo + RDV | | |

Programming Notes: Include randomized subjects only. Sort Order = Treatment Group, Disease Severity, USUBJID.

**Listing 2:** Subjects who Early Terminated or Discontinued Treatment

| Actual Treatment Group | Actual Disease<br>Severity | Subject ID | Category | Treatment Discontinued | Reason for Early Termination or Treatment<br>Discontinuation | Study Day |
|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate /<br>Severe | XXXXX | Early Termination/Treatment Discontinuation | NA/Infusions/Tablets/Infusions +<br>Tablets | Xxxxxx | xxxx |

Programming Notes: Sort Order = Treatment Group, Actual Severity, USUBJID, category where Treatment discontinuation is sorted prior to Early termination. If there are multiple treatment discontinuations (i.e. distinct dates for each product type) the order will be sorted by Study day. If both treatments were discontinued at the same time "Infusions + Tablets" will be displayed in the Treatment Discontinued column. If subjects were randomized and not dosed are categorized as "Not Treated" and sorted after Placebo + RDV if applicable.

**Listing 3:** Subject-Specific Protocol Deviations

| Actual Treatment<br>Group | Actual<br>Disease<br>Severity | Subject ID | DV Number | Deviation | Major/Minor<br>Designation | Deviation<br>Category | Study<br>Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/ | Moderate / | | | | | | | | | | | |
| Placebo + RDV | Severe | Xxxxx | XX | XXX | Major/Minor | XXX | X | xxxx | Yes/No | Yes/No | Yes/No | XXXX |

Programming Notes: Sort Order = Treatment Group, Actual severity, USUBJID, Deviation Number. Concatenate all the specify fields as appropriate. If the columns do not fit within the eCTD specified margins, then Actual Treatment Group, Actual Disease Severity, Subject ID will be placed in a header row as in the AE listings.

#### **Listing 4:** Non-Subject-Specific Protocol Deviations

| Site | Start Date | End Date | Deviation | Major/Minor<br>Designation | Reason for Deviation | Deviation Resulted in Subject Termination? | Deviation Affected<br>Product Stability? | Deviation<br>Category | Comments |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | XXXX | xxxx | Major/Minor | XXXX | Yes/No | Yes/No | XXXX | Xxxxx |

Programming Notes: Sort Order = Site (use site name and not the 5 alphanumeric site code), start date, deviation. Concatenate all the specify fields as appropriate

#### **Listing 5:** Individual Efficacy Response Data: Clinical Status Score Data

| Actual Treatment Group | Actual Disease Severity | Subject ID | Study Visit Day of Assessment | Actual Study Day of Assessment | Clinical Status Score | Clinical Status |
|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate / Severe | xxxxx | xx | xx | xx | xxxxx |

Programming Notes: Sort Order = Treatment Group, Actual severity, USUBJID, Study Day. Clinical status should match the wording of the scale definitions in Section 4.3.

**Listing 6: Individual Efficacy Response Data: NEWS** 

| Study Visit | Actual Study Respiratory Rate | | y Rate | O <sub>2</sub> Saturation | | Any Supplemental O <sub>2</sub> | | Temperature | | Systolic BP | | Heart Rate | | Level of<br>Consciousness | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | Day | bpm | Score | % | Score | Yes/No | Score | °C | Score | mmHg | Score | bpm | Score | A/V/P/U | Score | Score |
| Actual Treatment Group: , Actual Disease Severity: , Subject ID: | | | | | | | | | | | | | | | | |
| XX | xx | XX | XX | XX | XX | xx | XX | XX | XX | xx | XX | XX | xx | xx | xx | XX |

If the subject was on ECMO, heart rate and respiratory rate is denoted with a "-" and score of 3. If the subject is ventilated, the respiratory rate is denoted with a "-" and a score of 3.

Programming Notes: Sort Order = Treatment Group, Actual Severity, USUBJID, Study Visit Day.

**Listing 7:** Demographic Data

| Actual Treatment<br>Group | Actual Disease<br>Severity | Subject ID | Geographic<br>Region | Sex | Age at<br>Enrollment<br>(years) | Ethnicity | Race | Duration of Symptoms<br>prior to Enrollment<br>(Days) | Weight (Kg) | Height<br>(Cm) | BMI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate /<br>Severe | xxxxx | xxx | XXX | Xx | xxx | xxx | xxx | xx | Xx | Xxx |

Programming Notes: Sort Order = Treatment Group, Actual severity, USUBJID.

**Listing 8: Pre-Existing and Concurrent Medical Conditions** 

| Actual<br>Treatment<br>Group | Actual<br>Disease<br>Severity | Subject<br>ID | History of DVT or PE | Major Surgery, Significant<br>Trauma, Long<br>Hospitalization within one<br>month of screening | Prolonged Immobility<br>within one month of<br>screening | Medical History<br>Number | Medical History<br>Term | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|
| Baricitinib + | Moderate/ | | | | | 01 | xxxxx | Xxxx | xxxx |
| RDV/<br>Placebo + RDV | Severe | Xxx001 | Yes/No/Unknown | Yes/No/Unknown | Yes/No/Unknown | 02 | xxxxx | Xxxx | xxxx |

Programming Notes: Sort Order = Treatment Group, Actual Severity, USUBJID, MH Number. Each subject will have one row per medical condition reported on the Medical History CRF. If the subject reported "no" they do not have that pre-existing condition, the condition is not present in the line listing. If there is not enough space to fit all columns within the eCTD specified margins, then Actual Treatment Group, Actual Disease Severity, and Subject ID can be displayed in a header row as in the AE listings.

**Listing 9:** Concomitant Medications

| Actual Treatment<br>Group | Actual<br>Disease<br>Severity | Subject<br>ID | Medication<br>Number | Medication | Medication<br>Start Day | Medication<br>End Day | Indication | Taken for an AE?<br>(AE Description;<br>Number) | Taken for a condition on<br>Medical History?<br>(MH Description; Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate/<br>Severe | xxx | xx | xxxx | X | X | xxxx | Yes/No | Yes/No | xxxx / xxxx |

Programming Notes: Sort Order = Treatment Group, Actual severity, USUBJID, CM number

Note: If medication started prior to enrollment and there is no date, then Medication Start Day = Prior to Enrollment

If medication is ongoing at end of study, the Medication End Day = Ongoing

**Listing 10:** Medications of Interest

| Actual Treatment<br>Group | Actual Disease<br>Severity | Subject<br>ID | Medication<br>Number | Medication | Medication<br>Start Day | Medication<br>End Day | Indication | Medication of Interest<br>Category | Medication of Interest<br>Subcategory |
|---|---|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate/<br>Severe | xxx | XX | xxxx | X | X | xxxx | xxxx | xxxx |

Programming Notes: Sort Order = Treatment Group, Actual severity, USUBJID, CM number

Note: If medication started prior to enrollment and there is no date, then Medication Start Day = Prior to Enrollment

If medication is ongoing at end of study, the Medication End Day = Ongoing

If the medication does not have an applicable subcategory, then display 'N/A'

**Listing 11:** Compliance Data

| | | In | ifusions | | Tab | olets | | |
|---|---|---|---|---|---|---|---|---|
| Dose<br>Number | Infusion<br>Administered? | Infusion Slowed or<br>Stopped? | Reason(s) for Slowed/Stopped Infusion | Volume Administered if<br>Stopped/Slowed (mL) | Number of Tablets<br>Administered | Tablet Administered Successfully? | Reason for<br>Missed Dose | Comments |
| Actual Trea | | | | | | | | |
| 1 | Yes/No | No/Yes (Slowed)/Yes<br>(Stopped) | Xxxxx / NA | Xxx | 2/1 | Yes/No | Xxx/NA | |
| 2 | Yes/No | No/Yes (Slowed)/Yes<br>(Stopped) | Xxxxx / NA | Xxx | 2/1 | Yes/No | Xxx/NA | |
| | | | ••• | | | | ••• | |

Programming Notes: Sort Order = Treatment Group, Actual severity, USUBJID. If columns do not fit within the eCTD specified margins, then Study Day of Discharge and Study Day of Death can be added to the header row after Subject ID.

**Listing 12:** Listing of Non-Serious Adverse Events

| Adverse<br>Event | Study Day | Duration | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Unanticipated<br>Problem | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued Due<br>to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Actual Treatment Group: Actual Disease Severity: , Subject ID: , AE Number: | | | | | | | | | | | |
| xxx | xx | X | xxx | Related/Not<br>Related | XXXX | Yes/No | xxx | Yes/No | xxxx | xxxx | xxxx |
| Comments: xx | XX | | | | | | | | | | |

**Listing 13: Listing of Related Adverse Events** 

| Adverse<br>Event | Study Day | Duration | Severity | Unanticipated<br>Problem | Action Taken with<br>Study Treatment | Subject Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ Class | MedDRA<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|---|
| Actual Treat | Actual Treatment Group: Actual Disease Severity: , Subject ID: , AE Number: | | | | | | | | |
| xxx | XX | Х | xxx | Yes/No | xxx | Yes/No | xxxx | xxxx | xxxx |

Comments: xxx

**Listing 14:** Listing of Non-Fatal Serious Adverse Events

| Event | Study<br>Day<br>atment | Duration Group: , A | No. of Days Post First Dose the Event Became Serious ctual Disease Sever | Reason<br>Reported<br>as an<br>SAE<br>ity: , Subject | Severity ID: , AE N | Relationship<br>to Study<br>Treatment<br>umber: | If Not<br>Related,<br>Alternative<br>Etiology | Unanticipated<br>Problem | Taken<br>with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | х | X | X | xxxxx | XXX | Related/Not<br>Related | xxxx | Yes/No | XXXX | Yes/No | xxxxx | xxxxx | xxxxx |

**Listing 15:** Listing of Infections

| Study Day | Anatomical Location | Pathogen 1 | Pathogen 2 | Pathogen 3 | Pathogen 4 | Associated with AE Number | Secondary AE Number |
|---|---|---|---|---|---|---|---|
| Actual Treats | nent Group: , Actual Dis | sease Severity: , Subje | ect ID: | | | | |
| xx | xxx | xxx | xxx | XXX | XXX | xxx | xxx |

Listing 16: **Listing of Deaths** 

| Adverse<br>Event | Study<br>Day | Duration | No. of Days Post<br>First Dose the<br>Event Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Unanticipated<br>Problem | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Actual Tre | eatment G | roup: , Actu | ual Disease Severity: , | Subject ID: , | AE Number: | | | | | | | |
| xxxx | x | X | х | Xxxxx | xxx | Related/Not<br>Related | xxxx | Yes/No | xxxx | Yes/No | xxxxx | xxxxx |
| Comments: | : xxxx | | | | | | | | | | | |

Programming Note: Sort by actual treatment group, actual severity, USUBJID.

### **Listing 17:** Pregnancy Reports – Maternal Information

| Actual<br>Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal Complications During Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

**Listing 18:** Pregnancy Reports – Gravida and Para

| | | | | | | Live B | Births | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Actual<br>Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |
| Baricitinib<br>+ RDV/ | | | | | | | | | | | | | | | | |
| Placebo +<br>RDV | | | | | | | | | | | | | | | | |

Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

**Listing 19:** Pregnancy Reports – Live Birth Outcomes

| Actual<br>Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month<br>of Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baricitinib<br>+ RDV/ | | | | | | | | | | | | | |
| Placebo + | | | | | | | | | | | | | |
| RDV | | | | | | | | | | | | | |
| G : 1.1 | 1' | | | . 1 | | | | | | | | | |

Congenital Anomalies are included in the Adverse Event listing.

## **Listing 20:** Pregnancy Reports – Still Birth Outcomes

| Actual<br>Treatment<br>Group | Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baricitinib<br>+ RDV/ | | | | | | | | | | | | |
| Placebo + | | | | | | | | | | | | |
| RDV | | | | | | | | | | | | |

# **Listing 21:** Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Actual<br>Treatment<br>Group | Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy<br>Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/ | | | | | | | |
| Placebo + RDV | | | | | | | |

**Listing 22: Clinical Laboratory Results** 

| Actual Treatment<br>Group | Actual<br>Disease<br>Severity | Subject ID | Planned<br>Time Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory<br>Parameter (Units) | Result<br>(Toxicity Grade) | Change from<br>Baseline | Reference<br>Range Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate/<br>Severe | xxx | xx | xx | Xx | x | xxx (xxx) | xxx (xxxx) | xxx | xxxx | xxxx |

Programming Note: Sort order will be treatment group, Actual severity, USUBJID, planned time point, and lab parameter. If subjects were randomized and not dosed "Not Treated" will be used for the actual treatment category and will be sorted after Placebo+ RDV. All parameters will be included in the listing.

**Listing 23: Physical Exam Findings** 

| Actual Treatment<br>Group | Actual Disease Severity | Subject ID | Planned<br>Study Day | Actual<br>Study Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|---|
| Baricitinib + RDV/<br>Placebo + RDV | Moderate/Severe | xxx | xx | xx | xxxx | xxxxxx | Yes/No/NA |

Programming Note: For respiratory findings denoted as 'Yes' on the Physical Exam CRF, denote the Body System as "Respiratory Finding' and denote the Abnormal Finding as the symptom name; e.g. if Wheezing is reported, the Abnormal Finding will be 'Wheezing'. The Reported as an AE cell will be denoted as 'NA' for respiratory findings. Each reported respiratory finding will appear in its own row. If the finding was not reported as an AE as recorded on the CRF or the site did not report whether the finding was reported as an AE, the cell will display 'No'.

Sort order will be treatment group, actual severity, USUBJID, planned time point, and body system.

**Listing 24:** Subjects who Received the Incorrect Treatment

| Subject ID | Randomized Treatment<br>Group | Number of Infusions<br>Received | Number of Doses Received | Number of Incorrect Doses<br>Received |
|---|---|---|---|---|
| xxx | Baricitinib + RDV/<br>Placebo + RDV | X | x | X |

#### **Listing 25:** Subjects Randomized to the Incorrect Disease Severity Stratum

| Subject ID | Actual Treatment Group | Randomized Disease Severity | Actual Disease Severity |
|---|---|---|---|
| xxx | Baricitinib + RDV/<br>Placebo + RDV | Moderate/Severe | Moderate/Severe |

Programming Note: Sort but USUBJID. If subjects were randomized and not dosed "Not Treated" will be used for the actual treatment category.